

# PM60184-A-003-14

Phase I Multicenter, Open-label, Clinical and Pharmacokinetic Study of PM060184 in Combination with Gemcitabine in Selected Patients with Advanced Solid Tumors

# STATISTICAL ANALYSIS PLAN

| Version | Date | Description |
|---------|-------------|-------------|
| V1 0 | 23-Dec-2014 | Version 1.0 |

# **Table of Contents**

| List of Abbreviations | 5 |
|---------------------------------------------------|----|
| 1. Introduction | 7 |
| 2. Study Objectives | 7 |
| 2.1. Primary Objective | 7 |
| | 7 |
| 3. Study Design | |
| 4. Sample Size and Dose Escalation | 8 |
| 4.1. Sample size | 8 |
| 4.2. Dose escalation schedule | 8 |
| 5. Population and Endpoints | 10 |
| 5.1. Patient evaluability criteria | 10 |
| 5.2. Replacement of patients | 11 |
| 5.3. Endpoints | 13 |
| 5.3.1. Primary endpoint | 12 |
| 5.3.2. Secondary endpoints | 14 |
| 6. General Analysis Methods | 15 |
| 6.1. Statistical software | 15 |
| 7. Statistical Analysis | 16 |
| 7.1. Patient disposition and protocol deviations | 16 |
| 7.2. Baseline characteristics | 17 |
| 7.2.1. Demographics | 17 |
| 7.3. Statistical analysis for safety | 18 |
| 7.3.1. Treatment administration | 19 |
| 7.3.1. Cycle delays | 20 |
| 7.3.1. Dose omissions | 20 |
| 7.3.2. Dose modifications | 20 |
| 7.3.1. Adverse events | 21 |
| 7.3.1. Serious adverse event (SAE) | 21 |
| 7.3.1. Laboratory evaluations | 22 |
| 7.3.1. Physical examination | 23 |
| 7.3.2. ECG / LVEF | 23 |
| 7.3.3. Vital signs | 23 |
| 7.3.4. Concomitant medication | 23 |
| 7.4. Statistical analysis for efficacy | 24 |
| 7.4.1. Exploratory analysis of antitumor activity | 24 |
| 7.4.2. Level of significance | 24 |
| 7.5. Pharmacokinetics | 24 |
| 8. Other Statistical Analysis | 24 |
| 8.1. Stratification and covariate analysis | 24 |
| 8.2. Multivariate analysis | 25 |

| 8.3. Su | bgroup analysis | 25 |
|---|---|---|
| 8.4. Int | terim analysis | 25 |
| 8.5. Mi | issing values management | 25 |
| | Imputation of incomplete dates | 25 |
| 9. Tables, | Listings And Figures | 26 |
| 10. Appe | endix I. Patients Disposition | 29 |
| 10.1. Ge | eneral characteristics | 29 |
| <u>10.1.1.</u> | Patients treated, eligible and evaluable | 29 |
| 10.1.2. | Treatment discontinuations | 30 |
| 10.1.3. | Protocol deviations | 31 |
| 10.2. Pa | tient characteristics | 31 |
| <u>10.2.1.</u> | Patient characteristics at baseline | 31 |
| <u>10.2.2.</u> | Cancer history | 32 |
| 10.2.3. | Sites involved | 33 |
| 10.2.4. | Previous treatment summary | 34 |
| 10.2.5. | Physical examination, vital signs, electrocardiogram and other tests | 35 |
| 10.2.6.<br>10.2.7. | Hematological evaluation at baseline Biochemical evaluation at baseline | 37<br>38 |
| 10.2.7.<br>10.2.8. | Signs and symptoms at baseline | 39 |
| 10.2.9. | Concomitant medication starting pre-study | 41 |
| <u> 1. Appe</u> | endix II. Safety Evaluation | 42 |
| | tent of exposure | 42 |
| 11.1.1. | · | 42 |
| <u>11.1.2.</u> | Cumulative Dose, Dose Intensity and Relative Dose Intensity: Gemcitabine | 43 |
| 11.1.3. | | 44 |
| <u>11.1.4.</u> | Cycle Delays: Gemcitabine Dose Omission: PM060184 | 46<br>47 |
| 11.1.5.<br>11.1.6. | Dose Omission: Gemcitabine | 48 |
| 11.1.7. | Dose Modification: PM060184 | 49 |
| 11.1.8. | Dose Modification: Gemcitabine | 50 |
| 11.2. Do | se-limiting toxicities (DLT) | 51 |
| 11.2.1. | | 51 |
| | <u> </u> | |
| 11.3. Au | Verse events (AEs) Display of adverse events | <b>52</b> |
| | aths and other serious adverse events | 56 |
| 11.4.1. | Deaths | 56 |
| <u>11.4.2.</u> | Serious adverse events | 57 |
| 11.5. Cl | inical laboratory evaluation | 61 |
| 11.5.1. | Hematological abnormalities | 61 |
| 11.5.2. | Biochemical abnormalities | 62 |
| 11.5.3. | Laboratory Values over Time | 63 |
| 11.6. Ot | her observation related to safety | 66 |
| 11.6.1. | * | 66 |
| 11.7. Co | encomitant medication | 71 |
| 11.7.1. | Concomitant medication during study | 71 |
| <u>12. Appe</u> | andix III. Efficacy Evaluation | 72 |
| <b>12.1.</b> Ef | ficacy analysis | 72 |

| 12.1.1. Response | 72 |
|-----------------------------|-----------|
| 13. Figures | 75 |
| 13.1. Hematological profile | _75 |
| 13.2. Transaminase Profile | 76 |
| 13.3. Time to event graphs | |
| 14. Database Listings | <i>79</i> |

#### LIST OF ABBREVIATIONS

**AE(s)** Adverse Event(s)

ALT Alanine Aminotransferase
ANC Absolute Neutrophil Count
AP Alkaline Phosphatase

**aPTT** Activated Plasma Thromboplastin Time

**AST** Aspartate Aminotransferase

**AUC** Area Under The Concentration vs. Time Curve

**BSA** Body Surface Area

CL Clearance

Cmax Maximum Plasma Concentration

**CR** Complete Response

d/D Day(s)

DI Dose Intensity
DL Dose level

DLT Dose-limiting Toxicity
ECG Electrocardiogram
ECHO Echocardiography

**ECOG** Eastern Cooperative Oncology Group

**e-CRF** Electronic Case Report Form

**EORTC** European Organization for Research and Treatment of Cancer

**EOT** End of Treatment

**FUP** Follow-up

GCIG Gynecologic Cancer Intergroup

GCP Good Clinical Practice
GGT Gamma-glutamyltransferase
GIST Gastrointestinal Stromal Tumor
hCG Human Chorionic Gonadotropin

**ICH** International Conference on Harmonization

IEC Independent Ethics Committees
IRB Institutional Review Board
i.v. Intravenous (intravenously)

**LVEF** Left Ventricular Ejection Fraction

ml Milliliter

MTD Maximum Tolerated Dose

MUGA Multiple Gated Acquisition Scan NCA Non-compartmental Analysis NCI National Cancer Institute

NCI-CTCAE

National Cancer Institute-Common Terminology Criteria for Adverse

Events Events

ORR Overall Response Rate
OS Overall Survival
PD Progressive Disease
PFS Progression-free Survival

PhV Pharmacovigilance
PK Pharmacokinetic(s)
PR Partial Response

PRE TT Pre-treatment
PS Performance Status
PT Prothrombin Time
q3wk Every Three Weeks
q4wk Every Four Weeks
RD Recommended Dose

**RECIST** Response Evaluation Criteria In Solid Tumors

**SAE(s)** Serious Adverse Event(s)

**SD** Stable Disease

SUSAR/SUA Suspected Unexpected Serious Adverse Reaction

**TTP** Time To Progression

Uk Unknown

ULN Upper Limit of NormalWBC White Blood Cells

WHO World Health Organization

wk/wks Week/weeks

WMA World Medical Association

#### 1. INTRODUCTION

This document (Statistical Analysis Plan) explains in detail the statistical analyses that will be carried out for the PharmaMar PM60184-A-003-14 study.

The analyses described in this Statistical Analysis Plan are based upon and supplement those described in the Clinical Trial Protocol, version 1.0 (dated 28-Jul-2014).

#### 2. STUDY OBJECTIVES

The Clinical Trial Protocol states the following:

#### 2.1. Primary Objective

• To determine the maximum tolerated dose (MTD) and the recommended dose (RD) of PM060184 in combination with gemcitabine in selected patients with advanced solid tumors.

### 2.2. Secondary Objectives

- To characterize the safety profile and feasibility of this combination in this study population.
- To characterize the pharmacokinetics (PK) of this combination and to detect major drug-drug PK interactions.
- To obtain preliminary information on the clinical antitumor activity of this combination.

#### 3. STUDY DESIGN

Prospective, open-label, dose-ranging, uncontrolled phase I study with escalating doses of PM060184 in combination with gemcitabine in selected patients with advanced solid tumors.

Following a classical 3+3 design, successive cohorts of patients will receive escalating doses of intravenous (i.v.) gemcitabine over 30 minutes, followed by i.v. PM060184 over 10 minutes on Day 1 and Day 8 every three weeks (q3wk), until the RD is reached. All evaluable patients within a dose level (DL) must be followed for at least one full cycle (i.e., three weeks) before dose escalation may proceed to the next DL.

The MTD will be the lowest DL explored during dose escalation at which more than one third of evaluable patients experienced a DLT during Cycle 1. The RD will be the highest DL explored at which less than one third of evaluable patients experienced a DLT during Cycle 1. Dose escalation will cease immediately once the MTD is reached. Intermediate DLs can be tested, if deemed appropriate upon the Sponsor's and Investigators' agreement.

At least nine evaluable patients will be treated in an expansion cohort at the RD in order to evaluate its tolerability and feasibility. The tumor type(s) and/or target subpopulations to be included once the RD has been defined will be chosen according to the preliminary efficacy observed among patients treated during dose escalation, and will be discussed and agreed between the Investigators and the Sponsor, as appropriate.

### 4. SAMPLE SIZE AND DOSE ESCALATION

#### 4.1. Sample size

The number of patients may vary depending both on the tolerability of PM060184 combined with gemcitabine and the number of dose levels required to identify the MTD. Approximately between six and 36 evaluable patients are planned to be included in this study.

#### 4.2. Dose escalation schedule

The starting dose (DL1) for gemcitabine will be 800 mg/m<sup>2</sup>. This corresponds to a dose intensity (DI) of 533.33 mg/m<sup>2</sup>/week, and is equivalent to 80% of the RD with this schedule. This is the minimal gemcitabine dose accepted in clinical practice.

The DL1 for PM060184 will be  $6.0~\text{mg/m}^2$ . This corresponds to a DI of  $4.0~\text{mg/m}^2/\text{week}$ , and is equivalent to 64% of the RD determined for PM060184 given as single agent with this schedule.

The dose escalation scheme will follow pre-defined dose levels, starting at DL1, as summarized in the following table:

| DL | No. of patients | Relative DI (%) of gemcitabine / PM060184 | Gemcitabine dose (mg/m²) on Day 1 and Day 8 q3wk | PM060184 dose<br>(mg/m²)<br>on Day 1 and Day 8<br>q3wk |
|---|---|---|---|---|
| DL-1 | 0-6 | 80/53 | 800 | 5.0 |
| DL1 | 3-6 | 80/64 | 800 | 6.0 |
| DL2 | 3-6 | 80/74 | 800 | 7.0 |
| DL3 | 3-6 | 100/74 | 1000 | 7.0 |
| DL4 and<br>beyond | 3-6 | | No further dose increases beyond 1000 mg/m <sup>2</sup> | Further dose increases of 0.5 or 1.0 mg/m <sup>2</sup> , according to observed toxicities |
| DI, dose inter | nsity; DL, do | se level; MTD, maxir | num tolerated dose. | |

- Cohorts of at least three fully evaluable patients will be treated at each cohort.
- The second and third patients of a cohort may be included simultaneously after the first patient has completed the first cycle, except if a DLT is reported in the first patient, in which case the third patient of the cohort will be included once the second patient has received a complete treatment cycle with no reported DLTs. All patients will have to be fully evaluable (3-week period) prior to any further dose escalation. Patients not fully evaluable will be replaced.
- Dose escalation will continue if no DLT is observed.
- Subsequent dose levels will enroll three patients, and up to six fully evaluable patients if one DLT is observed in any of the first three fully evaluable patients.
- Once a DLT is observed, further patients will be included up to six fully evaluable patients in this dose cohort.

| No. of patients evaluable for DLT | No. of patients with DLTs in Cycle 1 | Action |
|---|---|---|
| 3 | 0 | Escalate DL |
| | 1 | Add 3 patients |
| | >1 | MTD |
| 6 | 1 | Escalate DL |
| | >1 | MTD |
| DL, dose level; DLT, dose | e-limiting toxicities; MTD, maximum to | olerated dose. |

- For gemcitabine: two doses (800 mg/m² and 1000 mg/m²) will be initially tested. If the toxicity observed during dose escalation is clearly related to gemcitabine (i.e. neutropenia and/or thrombocytopenia), intermediate gemcitabine doses might be tested after agreement between the Investigators and the Sponsor.
- For PM060184: pre-established PM060184 doses have been set for the first three DLs. After DL3, dose increments of 1.0 mg/m² will be tested if toxicity at each previous DL is acceptable. These dose increments may be of 0.5 mg/m², according to the toxicity observed. In the event of toxicities specifically related with PM060184 (i.e. peripheral neuropathy, post-infusion abdominal pain and/or diarrhea), intermediate PM060184 doses might be tested after agreement between the Investigators and the Sponsor.

Both the PM060184 and the gemcitabine doses may be rounded to the first decimal.

If more than one of three or six evaluable patients at any DL experience a DLT during Cycle 1, dose escalation will be terminated. The MTD will be the lowest level at which more than one third of evaluable patients experienced a DLT in Cycle 1. The RD will be the highest DL explored with less than one third of evaluable patients experiencing a DLT during Cycle 1.

If two or more evaluable patients (of 3-6 patients) at any DL experience a dose delay > 7 (+1) days from the theoretical due date (conforming or not to DLT criteria) and/or dose omissions exclusively related to PM060184 toxicity during Cycle 1, the cohort should be expanded as shown in the table below. If more than 50% of evaluable patients in a cohort experience dose delays and/or omissions, dose escalation will be terminated and this DL will be considered the MTD. An alternative schedule could then be explored after discussion between the Investigators and with the Sponsor's agreement. The starting dose of the new schedule will be the DL immediately below the MTD.

| Dose delays | Dose omissions | Action |
|---|---|---|
| 1 | - | None |
| - | 1 | None |
| 1 | 1 | Add 3 more patients |
| $\geq 2$ | - | Add 3 more patients |
| - | $\geq 2$ | Add 3 more patients |
| If more than 50% evaluable patient | s in a cohort have dose delays and/or | MTD |
| omissions | | |
| DLT, dose-limiting toxicities; MTD | , maximum tolerated dose. | |

An expansion cohort of a minimum of nine evaluable patients will be treated at the RD once it has been determined; this is to confirm its feasibility and tolerability. The tumor type(s) and/or target subpopulations that will be eligible to be included in this expansion cohort will be chosen according to the preliminary efficacy observed among those previously treated during dose escalation, and will be discussed and agreed between the Investigators and the Sponsor.

Intra-patient dose escalation will not be allowed under any circumstances.

### 5. POPULATION AND ENDPOINTS

Patients must fulfill all the inclusion/exclusion criteria to be eligible for admission to the study. See Clinical Trial Protocol, sections 4.1 Inclusion Criteria and 4.2 Exclusion Criteria

#### 5.1. Patient evaluability criteria

Analysis sets definitions:

"All Included Patients": it is defined as all patients who are included in the trial, independently of whether they have received the study drugs or not, excluding screen failure patients (Potential patient who did not meet one or more criteria at screening that was required for participation in the study).

All Evaluable Patients for the Assessment of the Primary Endpoint": A patient evaluable for the primary endpoint should have received at least one complete cycle (including the observation period). Patients who are discontinued early or miss/delay doses and/or assessments will be evaluable if these events are the consequence of treatment-related toxicity (excluding hypersensitivity reactions and/or extravasations).

"All Treated Patients (safety)":it is defined as all included patients who have received at least part of one infusion of PM060184/Gemcitabine.

"All Evaluable for Efficacy Patients": although it is not the main objective of this study, antitumor activity will be evaluated according to the RECIST v.1.1 in all patients with measurable disease, according to Choi criteria and/or EORTC metabolic response criteria for solid tumors in GIST patients, or by evaluation of serum tumor markers if applicable (e.g., ovarian cancer) every two cycles (i.e., approximately every six weeks) ± one week after treatment initiation until Cycle 4. Patients continuing treatment after Cycle 4 will have the assessments performed every three cycles (i.e., approximately every nine weeks) ± one week from Cycle 4 while on treatment, unless otherwise is clinically indicated. Patients included in the expansion cohort at the RD must be evaluable as per RECIST v.1.1 (or Choi criteria and/or EORTC metabolic response criteria for solid tumors, in the case of GIST), or by tumor markers

All analyses will be based on the actual treatment received by each patient rather than by the intended treatment. Any departures from the planned treatment according to the study schedule will be listed and documented in the clinical study report.

### 5.2. Replacement of patients

Patients must be replaced if they are not evaluable for the assessment of the primary endpoint, i.e. if:

- They are withdrawn from the study before receiving at least one evaluable cycle for any reason other than treatment-related toxicity (excluding hypersensitivity and/or extravasations reactions). An evaluable cycle is defined as: gemcitabine followed by PM060184 on Day 1 and Day 8, with the corresponding 2-week observation period during the first cycle.
- They require RT or other therapeutic procedure within three weeks after the first study drug dose, unless they previously had another treatment-related AE included in the definition of DLT.

• There is a protocol violation resulting in an impossibility of concluding anything regarding the safety of the study therapy.

All replaced patients will be included in the general safety analysis and in the efficacy analysis (if appropriate).

### 5.3. Endpoints

#### 5.3.1. Primary endpoint

#### **5.3.1.1.** Determination of MTD and RD

The MTD will be the lowest DL explored during dose escalation at which more than one third of evaluable patients experienced a DLT during Cycle 1.

The RD will be the highest DL explored at which less than one third of evaluable patients experience a DLT during Cycle 1. This RD will be confirmed if less than one third of the first nine evaluable patients treated during expansion have DLTs during their Cycle 1.

A patient evaluable for the primary endpoint should have received at least one complete cycle (including the observation period). Patients who are discontinued early or miss/delay doses and/or assessments will be evaluable if these events are the consequence of treatment-related toxicity (excluding hypersensitivity reactions and/or extravasations).

#### 5.3.1.2. DLT criteria

DLTs are defined as AEs and laboratory abnormalities related to the study treatment that occurred during Cycle 1 and fulfilled at least one of the following criteria:

- Grade 4 neutropenia (ANC  $< 0.5 \times 10^9/I$ ) lasting > 3 days.
- Grade  $\geq$  3 febrile neutropenia of any duration or neutropenic sepsis.
- Grade 4 thrombocytopenia (platelet count  $< 25 \times 10^9$ /l) or grade 3 with any major bleeding episode requiring a platelet transfusion.
- Grade 4 ALT and/or AST increase, or grade 3 lasting > 7 days.
- Treatment-related grade  $\geq 2$  ALT or AST increase concomitantly with  $\geq 2$  x ULN total bilirubin increase and normal AP.
- Any other grade 3/4 non-hematological AE that is suspected to be related to study drug(s), except nausea/vomiting (unless the patient is receiving an optimal antiemetic regimen), hypersensitivity reactions, extravasations, grade 3 asthenia lasting less than one week, anorexia, and non-clinically relevant isolated biochemical abnormalities [e.g., isolated increase in gamma-glutamyltransferase (GGT)]. In any case, the clinical relevance should be discussed between the Investigators and the Sponsor's representatives.

• Delay in the administration of Cycle 2 of the combination exceeding seven (+1) days of the treatment due date (i.e., Day 22), due to any AEs related to study drug(s).

The following circumstances will be discussed between the Principal Investigator and the Sponsor, and the final consensus will be documented:

- ✓ DLTs with delayed onset (i.e., that occur after Cycle 1).
- Non-compliance with the intended dose intensity (DI) in more than half of patients at any dose level (i.e., missing infusions on Day 8 or frequent dose delays due to treatment-related toxicity despite not conforming to a formal DLT definition).

### **5.3.2. Secondary endpoints**

- <u>Safety:</u> patients will be evaluable for safety if they have received at least one partial or complete infusion of PM060184 and one partial or complete infusion of gemcitabine. AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.4.
- **Pharmacokinetics:** PK analyses will be evaluated in plasma by standard non-compartmental analysis (NCA) (compartmental modeling may be performed if appropriate).
- <u>Pharmacogenetics:</u> a blood sample will be collected to evaluate the presence or absence of known polymorphisms that may explain individual variability in main PK parameters.
- Efficacy: although it is not the main objective of this study, antitumor activity will be evaluated according to RECIST v.1.1 in all patients with measurable disease, according to Choi criteria and/or EORTC metabolic response criteria for solid tumors, in GIST patients, or by evaluation of serum tumor markers if applicable (e.g., ovarian cancer), every two cycles (i.e., approximately every six weeks) ± one week after treatment initiation until Cycle 4. Patients continuing treatment after Cycle 4 will have the assessments performed every three cycles (i.e., approximately every nine weeks) ± one week from Cycle 4 while on treatment, unless otherwise is clinically indicated. Patients included in the expansion cohort at the RD must be evaluable as per RECIST v.1.1 (or Choi criteria and/or EORTC metabolic response criteria for solid tumors, in GIST patients) or by tumor markers.

Safety endpoints include:

- Adverse events (AEs).
- Hematology.
- Clinical chemistry.
- Coagulation tests.
- Vital signs.

- ECG and LVEF.
- Physical examinations.

Efficacy endpoints include:

Best overall response: defined as the best response achieved during the study according to RECIST / GCIG (ovarian cancer) / Choi criteria and/or EORTC metabolic response criteria for solid tumors (GIST), before disease progression, administration of subsequent anticancer treatment or study discontinuation.

Response rate (RR): defined as the ratio of patients with any response (CR or PR) divided by the total number of patients included in the efficacy population. The number of patients with  $SD \ge 4$  months will also be shown.

Duration of overall response: calculated from the date of first documentation of response (CR or PR, whichever comes first) to the date of documented PD or death. The censoring rules defined for PFS will be used for duration of response.

Progression-free survival: calculated as the time from the date of first drug administration to the date of documented progression or death (regardless of the cause of death). If the patient receives further antitumor therapy or is lost to follow-up before PD, PFS will be censored at the date of last tumor assessment before the date of subsequent antitumor treatment.

In patients with disease evaluable by serum markers, tumor assessments will be obtained every two cycles (i.e., every six weeks) and tumor response will be evaluated by GCIG specific criteria in patients with ovarian cancer. (see details in study protocol, Appendices 3 and 6).

#### 6. GENERAL ANALYSIS METHODS

#### 6.1. Statistical software

Medidata Rave® electronic data capture (EDC) will be used for data entry and clinical data management. SAS® Software v9.2 (or above) will be used for all statistical analyses.

#### 7. STATISTICAL ANALYSIS

### 7.1. Patient disposition and protocol deviations

Patients and dose levels will be summarized and listed by the populations used in the study:

- All included patients.
- All treated patients.
- All patients evaluable for the primary endpoint.
- All patients evaluable for efficacy.

Reasons for not belonging to any of these populations will be detailed.

The accrual and study discontinuation details will be presented descriptively.

Reasons for treatment discontinuation by number of cycles received will be described by counts and percentages. Reasons for treatment discontinuation other than disease progression will be detailed.

A protocol deviation is defined as any departure from what is described in the protocol of a clinical trial approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) and Competent Authorities. Therefore, it applies to deviations related to patient inclusion and clinical procedures (e.g., assessments to be conducted or parameters to be determined), and also to other procedures described in the protocol that concern the Good Clinical Practice (GCP) guidelines or ethical issues (e.g., issues related to obtaining the patients' Informed Consent, data reporting, the responsibilities of the Investigator, etc.).

Protocol deviations will be categorized by the Sponsor's responsible physician and summarized for all patients. A summary table with the number of patients with inclusion/exclusion deviations will be presented per criterion. These patients will be listed with the unmet criterion. Deviations with no effects on the risk/benefit ratio of the clinical trial (such as minimal delays in assessments or visits) will be distinguished from those that might have an effect on this risk/benefit ratio.

A summary including, but not necessarily restricted to, the following categories will be presented:

- Ineligible patients as per protocol.
- Patients not withdrawn as per protocol.
- Excluded concomitant medications.
- Incorrect dose or schedule, including patients not meeting re-treatment criteria on Day 1 and 8 of subsequent cycles.
- Failure to comply with study procedures.

#### 7.2. Baseline characteristics

#### 7.2.1. Demographics

Demographics and baseline characteristics will be summarized for all patients. All subject characteristics descriptions will be performed by dose level (or most adequate dose grouping).

Continuous variables will be summarized and presented with summary statistics, i.e., mean, median, range and standard deviation.

Categorical variables will be summarized in frequency tables. Percentages in the summary tables will be rounded and may therefore not always add up to exactly 100%.

In case of pre-treatment characteristics with multiple measurements per patient before the start of treatment (laboratory assessments, vital signs), the baseline measurement will be considered the last value prior to or on the first day of treatment.

Baseline BSA will be calculated using the Dubois & Dubois formula:

$$BSA(m^2) = 0.007184 \times weight(kg)^{0.425} \times height(cm)^{0.725}$$

Age will be calculated based on the date of birth and the date of informed consent. Age categories and race will be summarized with frequency counts.

$$Age = \frac{\text{(date of informed consent) - (date of birth)}}{365.25}$$

Baseline body mass index (BMI) will be calculated, using the formula:

$$BMI = \frac{weight(kg)}{height(m)^2}$$

Baseline ECOG will be summarized with frequency counts.

For cancer history, histological diagnosis, time from diagnosis, number of baseline lesions, and involvement in the different sites will be summarized. Time from initial diagnosis to the start of current treatment and time from the latest disease progression to the start of current treatment will be calculated in months and summarized descriptively. If incomplete dates are recorded, rules described in section <u>8.5</u> will be used for imputation.

Primary tumor sites and baseline lesions will be recoded by the Sponsor's physicians to categorize them accurately in the analysis.

Previous relevant medical history (other than cancer) will be listed by dose level (or most adequate dose grouping) and patient.

A frequency tabulation of the different types of previous cancer surgery, radiotherapy, or anticancer systemic therapy (number of lines and number of agents) will be given. Chemotherapy agents and lines will be recoded by the Sponsor's physicians to categorize them accurately in the analysis.

Signs and symptoms, hematology and serum biochemistry abnormalities at baseline will be displayed by tabulation of frequencies according to NCI-CTCAE v4.03 toxicity grades. Signs and symptoms and laboratory abnormalities of grade  $\geq 2$  at baseline will be listed by dose level (or most adequate dose grouping) and patient.

#### 7.3. Statistical analysis for safety

All analyses of safety variables will be descriptive. Data retrieved at both scheduled and unscheduled visits will be tabulated and listed.

The safety population consists of all patients who receive at least part of a PM060184/Gemcitabine infusion. The safety patient population will be used for the general safety presentations.

In particular, for the evaluation of the primary endpoint, the total number of patients included, the number of patients evaluable for determination of DLTs, and the number of patients with any DLT (and their categorization) will be summarized by dose level (or most adequate dose grouping). The toxicities meeting the DLT criteria in Cycle 1 and subsequent cycles, if any, will be listed separately, and the description of laboratory abnormalities (hematology/biochemistry) will be supported by graphs depicting the evolution in time of laboratory values (including nadir calculation and median time to recovery from baseline values).

#### 7.3.1. Treatment administration

<u>Exposure to treatment</u> will be described by dose level for all patients who have received at least one of the study drugs.

<u>Total cumulative dose</u>, expressed in mg  $/m^2$ , is the sum of all the product doses from Cycle 1 until the dose received in the last cycle.

<u>Intended dose intensity</u> is the planned dose for the cycle divided by the planned duration of a cycle in weeks.

Absolute dose intensity is the total cumulative dose divided by the duration of the treatment. As a convention, the duration of the last cycle is considered to be 21 days (planed cycle duration) even if the patient dies or receives another anticancer therapy before the end of the cycle.

<u>Relative dose intensity (%)</u> is the ratio of absolute dose intensity divided by the intended dose intensity.

<u>Time on treatment</u> is the distance, expressed in weeks, between the first infusion date and the last infusion date plus 30 days or start of new treatment or date of death (whichever occurs first).

The number of cases, median, standard deviations, minimum and maximum values for the parameters defined above will be tabulated by dose level (or most adequate dose grouping).

### 7.3.1. Cycle delays

The item "Infusion skipped/delayed: No/Yes" in the E-CRF will be used to calculate the delay. For doses considered as delayed by the Investigator, the delay will be calculated as:

Delay (in days) will be equal to the date of start of current cycle minus the date of start of previous cycle minus 21 days (planed cycle duration, in days).

The first cycle is excluded from all calculation of cycle delay (and the denominator used for calculations will be equal to the number of cycles susceptible to be delayed).

A second analysis taking into account the drug administration dates rather than the item "dose delay" completed by the Investigator will be performed in order to know the calculated delay in days.

The distribution of delays according to the infusion administered will be studied by means of counts and percentages. The reasons for infusion delay will be detailed, specifying how many were due to treatment and how many were not. Within delays attributable to treatment, hematological and non-hematological reasons will be outlined, and the specific reasons will be detailed (administrative reasons will be analyzed separately and additional tables will be prepared after exclusion of those delays).

#### 7.3.1. Dose omissions

Infusions not administered on Day 8 of a cycle will be considered skipped doses.

The distribution of omissions will be studied by means of counts and percentages. The reasons for infusion omission will be detailed, specifying how many were due to treatment and how many were not. Within omissions attributable to treatment, hematological and non-hematological reasons will be outlined, and the specific reasons will be detailed.

#### 7.3.2. Dose modifications

All dose reductions will be considered and described (per cycle and patient), specifying the magnitude and the reason for reduction (hematological toxicity, non-hematological toxicity or other causes not due to treatment).

#### 7.3.1. Adverse events

Toxicity will be evaluated according to the NCI-CTCAE v4.03 and the events will be coded and classified using the MedDRA dictionary.

As far as all the toxicities are concerned, the NCI-CTCAE grade will be used wherever an NCI-CTCAE grading exists. Otherwise, the severity will be noted. As a convention, the term "Grade" will always be used. Toxicities will be described according to the worst NCI-CTCAE grade or, for toxicities which do not form the subject of NCI-CTCAE classification, according to the worst severity.

Descriptive statistics will be used for the evaluation of safety. The incidence and grade of adverse events and laboratory abnormalities will be calculated considering the most severe grade per patient and infusion and will be displayed in frequency tables using counts and percentages.

The shift of severity grades from baseline to the worst occurrence during treatment will be tabulated.

Deaths, serious adverse events and events resulting in study discontinuation will be tabulated.

Additional safety analyses may be determined at any time, in order to most clearly enumerate rates of toxicities and to further define the safety profile of PM060184. In order to categorize accurately the safety information, additional classifications other than SOC/PT could be populated in order to understand better the safety drug profile.

#### 7.3.1. Serious adverse event (SAE)

Database listings of deaths and serious adverse events will be provided, including at least date of onset and resolution (if applicable), severity, relationship to study drug, most important significant consequence and main action taken.

### 7.3.1. Laboratory evaluations

#### 7.3.1.1. Hematology

Hematological toxicities classified according to the NCI-CTCAE v4.03 will be calculated in all cycles by dose level (or most adequate dose grouping). Separate analyses will be carried out for Cycle 1. The worst grade reached by each patient during treatment and Cycle 1 will also be calculated.

If serious toxicities occur, special follow-up including calculation of median and range of nadir values and median time to recover to baseline values and descriptive tables will be made to find out the pattern of thrombocytopenia and neutropenia within and between the different cycles.

If appropriate, these tables might be complemented with boxplots for the nadir of neutrophils and platelets count by cycle along the treatment by dose level (or most adequate dose grouping). Furthermore, graphs of the inter-cycle time course of neutropenia, thrombocytopenia or any other considered parameter will be provided. Eventually, graphs comparing the time course during the first and second cycles will be created.

#### 7.3.1.2. Serum biochemistry and coagulation tests

The non-hematological laboratory abnormalities (i.e. NCI-CTCAE grades) of transaminases, creatinine, creatine phosphokinase (CPK), bilirubin, alkaline phosphatase, etc. by patient and cycle will be calculated as explained for hematological toxicities. Separate analyses will be carried out for Cycle 1. The worst grade reached by each patient during treatment and Cycle 1 will also be calculated.

If serious toxicities occur, special follow-up including calculation of median and range of peak values and median time to recover to baseline values and descriptive tables will be made to find out the pattern of the involved toxicities within and between the different cycles.

If appropriate, these tables might be complemented with boxplots for the peaks of transaminases, creatinine, CPK, bilirubin, AP, etc. by cycle along the treatment by dose level (or most adequate dose grouping). Furthermore, graphs of the inter-cycle time course of any considered parameter will be provided. Eventually, graphs comparing the time course during the first and second cycles will be created.

### 7.3.1. Physical examination

The results of the physical examination (normal/abnormal) will be summarized with frequency counts. All data will be listed by dose level.

#### **7.3.2.** ECG / LVEF

The results of the baseline ECG evaluation (normal/abnormal) will be summarized with frequency counts.

Continuous variables (PR Interval, QT Interval, QRS Complex, Ventricular Rate, QTc (Fridericia's), LVEF and LVEF Normal Range) will be summarized and presented with summary statistics, i.e., mean, standard deviation, median and range. Tabulation of baseline values and evolution during treatment will be presented with summary statistics.

$$QTcF = \frac{QT}{\sqrt[3]{\frac{60}{\text{HR}}}}$$

HR = Heart Rate

QTc (Fridericia's) will be graded using NCI-CTCAE v4.03.

#### 7.3.3. Vital signs

Performance status and weight gain/loss during the study will be summarized by frequency tabulation.

#### 7.3.4. Concomitant medication

Concomitant therapies will be coded using WHO-ATC dictionary and categorized per ATC (levels 1, 2 and 4) class. The number of patients receiving each type of therapy will be tabulated in two separated tables: a frequency tabulation of the therapies that started before the study, and a frequency tabulation of those that started during the study. The accompanying listing will contain all concomitant therapies.

Additional listings for patients taking medications / therapies that were prohibited by protocol will be provided.

### 7.4. Statistical analysis for efficacy

### 7.4.1. Exploratory analysis of antitumor activity

Response rates as per RECIST v1.1 (and as per Choi criteria or EORTC metabolic response criteria for ovarian cancer and GIST patients, respectively) [percentage of patients with any response [PR, CR or the sum of both being the overall response rate (ORR)], percentage of patients with clinical benefit [i.e., patients with any response, or with stable disease  $(SD) \ge 4$  months], will be characterized using descriptive statistics (95%) exact binomial confidence interval) and according to primary tumor type. Time-related parameters (e.g., PFS) will also be analyzed according to the Kaplan-Meier method, if appropriate. If any specific tumor type subset is adequately represented, exploratory subgroup analyses will be performed. The characteristics of the patients achieving an objective response or  $SD \ge 4$  months by RECIST v1.1 will be displayed.

### 7.4.2. Level of significance

Confidence intervals will be constructed using the 95% level. No formal statistical tests are defined, but if needed, all will be done at a significance level of 5% and will be considered exploratory.

#### 7.5. Pharmacokinetics

Methods used and results will be provided in a separate document prepared by the Clinical Pharmacology department.

#### 8. OTHER STATISTICAL ANALYSIS

#### 8.1. Stratification and covariate analysis

No stratification by prognostic factors or tumor types is planned. If a disease is adequately represented, response rates might be analyzed descriptively, and time-related parameters might be analyzed according to the Kaplan-Meier method. Efficacy parameters could also be subjected to further appropriate analysis, considering correlation with factors of probable prognostic value such as patient PS at entry, stage of disease (locally advanced / metastatic stage), prior therapies, etc. using the appropriate test (Fisher's exact test, Spearman test, etc.).

#### 8.2. Multivariate analysis

If appropriate, exploratory *Cox* regression for multivariate analysis will be used for time-dependent efficacy parameters, and logistic regression for the evaluation of covariates associated with best overall response.

#### 8.3. Subgroup analysis

If ovarian and GIST cancer groups of patients are sufficiently represented, a separate analysis by tumor type and evaluation criteria (RECIST, GCIG, Choi) will be performed.

#### 8.4. Interim analysis

The patient's safety will be assessed on a regular basis prior to each dose escalation upon completion of a cohort. No formal interim analyses are planned.

### 8.5. Missing values management

Missing laboratory values will be subtracted from the tables.

#### 8.5.1. Imputation of incomplete dates

#### Dates before randomization

If day of a date is unknown then the imputed day will be 15, if the month is also unknown then the imputed date will be 01/July/year. This assumption will be valid if the imputed date is earlier than the informed consent's date; otherwise the imputed date will be the first day of the informed consent's month date (i.e. 01/ informed consent's month date/year).

### Dates after end of treatment

To ensure the most conservative approach for the main time-to-event variables (i.e., PFS) that can be affected by missing values, the following rules will be implemented: if the day of a date is unknown, then the imputed day will be 01; if the month is also unknown, then the imputed date will be 01/July/year. This assumption will be valid if the imputed date occurs later than the last drug administration date; otherwise, the imputed date will be the last drug administration date plus the planed cycle duration (21 days) or the last day of the reported month, whichever occurs first.

# 9. TABLES, LISTINGS AND FIGURES

All summary tables will have source data footnotes that refer to the relevant listings. All listings will be ordered by treatment (dosing, etc.), patient and cycle number.

| <i>Table 10.1.1.1</i> | Patient accrual by Institution and dose level | <b>2</b> 9 |
|---|---|---|
| <i>Table 10.1.1. 2</i> | Disposition of patients | 29 |
| <i>Table 10.1.1. 3</i> | Time on treatment by dose level | 29 |
| <i>Table 10.1.1. 4</i> | Number of patients evaluable for analysis | 29 |
| <i>Table 10.1.1. 5</i> | Number of patients evaluable for analysis | 29 |
| <i>Table 10.1.2. 1</i> | Treatment discontinuation by dose level | 30 |
| <i>Table 10.1.2. 2</i> | Treatment discontinuation details | 30 |
| <i>Table 10.1.2. 3</i> | Treatment discontinuation due to adverse events | 30 |
| <i>Table 10.1.2. 4</i> | Reasons for treatment discontinuation other than progressive disease | 30 |
| Table 10.1.2. 5 | Reasons for study discontinuation by dose level | 30 |
| Table 10.1.3. 1 | Protocol deviations | 31 |
| Table 10.2.1. 1 | Age at entry by dose level | 31 |
| Table 10.2.1. 2 | Supportive listing: Baseline demographics characteristic | 31 |
| Table 10.2.2. 1 | Primary tumor by dose level | 32 |
| Table 10.2.2. 2 | Prior cancer history time differences | 32 |
| Table 10.2.2. 3 | Other cancer history characteristics | 32 |
| Table 10.2.3. 1 | Supporting listing: Evaluation method | 33 |
| Table 10.2.3. 2 | Supportive listing: Sites of disease (RECIST v1.1) | 33 |
| Table 10.2.4. 1 | Previous treatment summary by dose level | 34 |
| Table 10.2.4. 2 | Previous surgery by dose level | 34 |
| Table 10.2.4. 3 | Previous radiotherapy by dose level | 34 |
| Table 10.2.4. 4 | Agents of previous anticancer therapies (ATC 1 & 4) by dose level | 34 |
| Table 10.2.4. 5 | No. of lines/agent of prior anticancer therapies by dose level | 35 |
| Table 10.2.5. 1 | Physical examination by dose level | 35 |
| Table 10.2.5. 2 | ECOG performance status by dose level | 36 |
| Table 10.2.5. 3 | Supportive listing: Patients with $PS \ge 2$ | 36 |
| Table 10.2.5. 4 | ECG by dose level | 36 |
| Table 10.2.5. 5 | LVEF by dose level | 37 |
| Table 10.2.5. 6 | Vital signs by dose level | 37 |
| Table 10.2.6. 1 | Hematological abnormalities by dose level | 37 |
| Table 10.2.6. 2 | Median and range for hematological parameters by dose level | 38 |
| Table 10.2.6. 3 | Supportive listing: Patients with grade ≥2 hematological abnormalities | 38 |
| Table 10.2.6. 4 | Supportive listing: Patients with missing grade for hematological abnormalities | 38 |
| Table 10.2.7. 1 | Biochemical abnormalities by dose level | 38 |
| Table 10.2.7. 2 | Median and range for biochemical parameters by dose level | 39 |
| Table 10.2.7. 3 | Supportive listing: Patients with grade ≥2 biochemical abnormalities | 39 |
| <i>Table 10.2.7. 4</i> | Supportive listing: Patients with missing grade for biochemical abnormalities | 39 |
| Table 10.2.8. 1 | Signs and symptoms by dose level | 39 |
| Table 10.2.8. 2 | Listing of grade ≥2 and not disease-related signs and symptoms | 39 |
| Table 10.2.8. 3 | Incidence of signs and symptoms by dose level | 41 |
| Table 10.2.9. 1 | Concomitant medication starting pre-study (ATC 1 and 4) by dose level | 41 |
| Table 10.2.9. 2 | Concomitant medication starting pre-study (Transfusions and/or EPO) | 41 |
| Table 10.2.9. 3 | Supportive listing: Patients with transfusions and/or EPO (pre-study) | 41 |
| Table 11.1.1. 1 | No. of cycles administered (PM060184) | 42 |
| Table 11.1.1. 2 | No. of cycles administered by dose level (PM060184) | 42 |
| Table 11.1.1. 3 | Cumulative dose, DI and RDI by dose level (PM060184) | 42 |
| Table 11.1.1. 4 | Supportive listing: Patients with less than 60% of RDI (PM060184) | 43 |
| Table 11.1.2. 1 | No. of cycles administered (gemcitabine) | 43 |
| Table 11.1.2. 2 | No. of cycles administered by dose level (gemcitabine) | 43 |
| Table 11.1.2. 3 | Cumulative dose, DI and RDI by dose level (gemcitabine) | 44 |

| <i>Table 11.1.2. 4</i> | Supportive listing: Patients with less than 60% of RDI (gemcitabine) | 44 |
|---|---|---|
| <i>Table 11.1.3. 1</i> | Summary of dose delay by dose level (PM060184) | 45 |
| <i>Table 11.1.3. 2</i> | Supportive listing: Dose delays (PM060184) | 45 |
| <i>Table 11.1.3. 3</i> | Supportive listing: Dose delays excluding administrative reasons (PM060184) | 45 |
| <i>Table 11.1.4.1</i> | Summary of dose delay by dose level (gemcitabine) | 46 |
| <i>Table 11.1.4. 2</i> | Supportive listing: Dose delays (gemcitabine) | 46 |
| Table 11.1.4. 3 | Supportive listing: Dose delays excluding administrative reasons (gemcitabine) | 46 |
| <i>Table 11.1.5. 1</i> | Summary of dose omission by dose level (PM060184) | 47 |
| Table 11.1.5. 2 | Listing of dose omissions (PM060184) | 47 |
| Table 11.1.6. 1 | Summary of dose omission by dose level (gemcitabine) | 48 |
| Table 11.1.6. 2 | Listing of dose omissions (gemcitabine) | 48 |
| Table 11.1.7. 1 | Summary of reduced cycles by dose level (PM060184) | 49 |
| Table 11.1.7. 2 | Listing of dose reductions (PM060184) | 49 |
| Table 11.1.8. 1 | Summary of reduced cycles by dose level (gemcitabine) | 50 |
| Table 11.1.8. 2 | Listing of dose reductions (gemcitabine) | 50 |
| Table 11.2.1. 1 | Summary of patients with DLT by dose level | 51 |
| Table 11.2.1. 2 | Details of DLT | 51 |
| Table 11.3.1. 1 | Drug-related (or relationship UK) AEs. Worst grade by patient | 52 |
| Table 11.3.1. 2 | Drug-related (or relationship UK) AEs in the first cycle | 52 |
| Table 11.3.1. 3 | Drug-related (or relationship UK) AEs. Worst grade per cycle | 52 |
| Table 11.3.1. 4 | Drug related (or relationship UK) AEs in $\geq 10\%$ of patients | 53 |
| Table 11.3.1. 5 | Drug related (or relationship UK) AEs in $\geq$ 10% of patients. Worst grade per cycl | |
| Table 11.3.1. 6 | AEs regardless of relationship. Worst grade by patient | 53 |
| Table 11.3.1. 7 | AEs regardless of relationship in the first cycle | 54 |
| <i>Table 11.3.1. 8</i> | AEs regardless of relationship. Worst grade per cycle | 54 |
| Table 11.3.1. 9 | AEs observed in ≥10% of cycles | 54 |
| Table 11.3.1. 10 | AEs observed in ≥10% of patients. Worst grade per cycle | 55 |
| Table 11.3.1. 11 | Supportive listing: Drug-related (or relationship UK) grade 2-4 AEs | 55 |
| Table 11.3.1. 12 | Supportive listing: All AEs regardless of relationship | 55 |
| Table 11.4.1. 1 | Patients who died while on treatment | 56 |
| Table 11.4.1. 2 | Patients who died within 30 days of last drug administration | 56 |
| Table 11.4.1. 3 | Listing of all deaths | 56 |
| Table 11.4.2. 1 | Drug-related (or relationship UK) SAEs. Worst grade by patient | 57 |
| Table 11.4.2. 2 | Drug-related (or relationship UK) SAEs in the first cycle | 57 |
| Table 11.4.2. 3 | Drug-related (or relationship UK) SAEs. Worst grade per cycle | 57 |
| Table 11.4.2. 4 | Drug related (or relationship UK) SAEs in ≥10% of patients | 58 |
| Table 11.4.2. 5 | Drug related (or relationship UK) SAEs in ≥10% of patients. Worst grade per cyc | |
| | 58 | |
| Table 11.4.2. 6 | SAEs regardless of relationship. Worst grade by patient | 58 |
| Table 11.4.2. 7 | SAEs regardless of relationship in the first cycle | 59 |
| <i>Table 11.4.2. 8</i> | SAEs regardless of relationship. Worst grade per cycle | 59 |
| <i>Table 11.4.2. 9</i> | SAEs observed in $\geq$ 10% of cycles | 59 |
| Table 11.4.2. 10 | SAEs observed in ≥10% of patients. Worst grade per cycle | 60 |
| Table 11.4.2. 11 | All SAEs | 60 |
| Table 11.5.1. 1 | Hematological abnormalities: Worst grade per patient | 61 |
| Table 11.5.1. 2 | Hematological abnormalities: Worst grade per cycle | 61 |
| Table 11.5.1. 3 | Supportive listing: Patients with grade ≥3 hematological abnormalities | 61 |
| Table 11.5.1. 4 | Supportive listing: Patients with missing grade for hematological abnormalities | 61 |
| Table 11.5.2. 1 | Biochemical abnormalities: Worst grade per patient | 62 |
| Table 11.5.2. 2 | Biochemical abnormalities: Worst grade per cycle | 62 |
| Table 11.5.2. 3 | Supportive listing: Patients with grade ≥3 biochemical abnormalities | 62 |
| Table 11.5.2. 4 | Supportive listing: Patients with missing grade for biochemical abnormalities | 62 |
| Table 11.5.3. 1 | Shift of hematological abnormalities. Baseline grade vs worst grade on treatment | |
| <i>Table 11.5.3. 2</i> | | |
| | Shift of biochemical abnormalities. Baseline grade vs worst grade on treatment | |
| Table 11.5.3. 3 | Shift of biochemical abnormalities. Baseline grade vs worst grade on treatment | 64 |
| | • | 64<br>65 |

| <i>Table 11.5.3. 5</i> | Pattern of neutropenia/thrombocytopenia | 65 |
|---|---|---|
| <i>Table 11.5.3. 6</i> | Pattern of hepatobiliary parameters | 65 |
| <i>Table 11.6.1. 1</i> | Performance status during the study by cycle and dose level | 66 |
| <i>Table 11.6.1. 2</i> | Physical examination during the study by cycle and dose level | 66 |
| <i>Table 11.6.1. 3</i> | Weight gain-loss during the study by dose level | 67 |
| <i>Table 11.6.1. 4</i> | Vital sign (pulse) during the study by cycle and dose level | 67 |
| <i>Table 11.6.1. 5</i> | Vital sign (temperature) during the study by cycle and dose level | 67 |
| <i>Table 11.6.1. 6</i> | Vital sign (BPS) during the study by cycle and dose level | 68 |
| <i>Table 11.6.1. 7</i> | Vital sign (BPD) during the study by cycle and dose level | 68 |
| <i>Table 11.6.1. 8</i> | ECG during the study by cycle and dose level | 68 |
| <i>Table 11.6.1. 9</i> | ECG (PRI) during the study by cycle and dose level | 69 |
| <i>Table 11.6.1. 10</i> | ECG (QTI) during the study by cycle and dose level | 69 |
| <i>Table 11.6.1. 11</i> | ECG (QTc) during the study by cycle and dose level | 69 |
| <i>Table 11.6.1. 12</i> | ECG (VR) during the study by cycle and dose level | 70 |
| <i>Table 11.7.1. 1</i> | Concomitant medication during study (ATC 1 and 4) by dose level | 71 |
| <i>Table 11.7.1. 2</i> | Transfusions / EPO (Patients with transfusions and/or EPO) | 71 |
| <i>Table 12.1.1. 1</i> | Overall response by dose level. Treated patients | 72 |
| <i>Table 12.1.1. 2</i> | Overall response by dose level. Evaluable patients | 72 |
| <i>Table 12.1.1. 3</i> | Tumor marker evolution during the study | 72 |
| <i>Table 12.1.1. 4</i> | Progression-free survival. Treated population | 73 |
| <i>Table 12.1.1. 5</i> | Progression-free survival. Evaluable population | 73 |
| <i>Table 12.1.1. 6</i> | Duration of response | 73 |
| <i>Table 12.1.1. 7</i> | Characteristics of patients with evidence of clinical benefit* | 74 |
| <i>Table 12.1.1. 8</i> | Supportive listing: efficacy dataset analyzed | 74 |
| Figure 13.1. 1 | Pattern of hematological/non-hematological DLTs in individual patients | 75 |
| Figure 13.2. 1 | Transaminase series. Patient XX | <del>76</del> |
| Figure 13.2. 2 | Bar charts of hematological/biochemical laboratory abnormalities by dose level | 76 |
| Figure 13.2. 3 | Hematology / Transaminase. Worst severity by cycle | 77 |
| Figure 13.3. 1 | Progression-free survival (PFS) | <i>78</i> |

### 10. APPENDIX I. PATIENTS DISPOSITION

#### 10.1. General characteristics

### 10.1.1. Patients treated, eligible and evaluable

Table 10.1.1. 1 Patient accrual by Institution and dose level

| Institution | DL1 | DL2 | DL3 | | Total |
|---------------|------|------|------|------|-------|
| | N(%) | N(%) | N(%) | N(%) | N(%) |
| Institution 1 | | | | | |
| Institution 2 | | | | | |

Note: Percentage is based on number of patients by dose level.

### Table 10.1.1. 2 Disposition of patients

| Dates information |
|------------------------------------|
| Date of first consent |
| Date of first dose |
| Date of last consent |
| Date of first dose of last patient |
| Date of last dose |
| Date of last follow up* |

(\*) Last follow up date, examination date or procedure before study closure.

Table 10.1.1. 3 Time on treatment by dose level

| Median and range of time on treatment (weeks) | DL1 | DL2 | DL3 | <br>Total |
|-----------------------------------------------|-----|-----|-----|-----------|
| N | | | | |
| Median (range) | | | | |
| Mean (std) | | | | |

Table 10.1.1.4 Number of patients evaluable for analysis

| | DL I | DL2 | DL3 | | Lotal |
|------------------------|------|------|------|------|-------|
| | N(%) | N(%) | N(%) | N(%) | N(%) |
| All included patients | | | | | |
| Evaluable for DLT | | | | | |
| Evaluable for safety | | | | | |
| Evaluable for efficacy | | | | | |

Table 10.1.1. 5 Number of patients evaluable for analysis

| Not evaluable for | Dose level | Patient | Reason(s) |
|---------------------------|------------|---------|-----------|
| DLT<br>Safety<br>Efficacy | | | |
| Safety | | | |
| Efficacy | | | |
| ••• | | | |

#### 10.1.2. Treatment discontinuations

Table 10.1.2. 1 Treatment discontinuation by dose level

| DL1 | DL2 | DL3 | | Total |
|------|------|------|------|-------|
| N(%) | N(%) | N(%) | N(%) | N(%) |

Progressive disease

Patient refusal

Death

Investigator's decision

Treatment-related adverse event

Non treatment-related adverse event

Other

Total

Notes: Percentage is based on number of patients by dose level.

Table 10.1.2. 2 Treatment discontinuation details

| Dose level | Patient No. | Last cycle infused | Treatment discontinuation reason | Details |
|---|---|---|---|---|

Table 10.1.2. 3 Treatment discontinuation due to adverse events

| Dose level | Patient No. | SOC/Group | PT/sub-group | Relationship |
|------------|-------------|-----------|--------------|--------------|

Table 10.1.2. 4 Reasons for treatment discontinuation other than progressive disease

| 14010 10.1.2. 1 | reasons re | or treatment disconti | naution other than pre | Gressive disease |
|---|---|---|---|---|
| Dose level | Patient No. | Last cycle infused | Off Study reason | Specify |

Table 10.1.2. 5 Reasons for study discontinuation by dose level

| DL1 | DL2 | DL3 | | Total |
|------|------|------|------|-------|
| N(%) | N(%) | N(%) | N(%) | N(%) |

Study termination (clinical cut-off)

Patient's follow-up completed

Patient's refusal

Death

Never treated

Lost to follow up

Other

Total

Note: Percentage is based on number of patients by dose level.

#### 10.1.3. Protocol deviations

### Table 10.1.3. 1 Protocol deviations

| Dose level | Patient No. | Protocol deviation type | Specify |
|------------|-------------|-------------------------|---------|

### 10.2. Patient characteristics

### 10.2.1. Patient characteristics at baseline

Table 10.2.1. 1 Age at entry by dose level

| | DL1 | DL2 | DL3 | | Total |
|----------------------|------|------|------|------|-------|
| | N(%) | N(%) | N(%) | N(%) | N(%) |
| Age at entry | | | | | |
| 18-XX years | | | | | |
| XX-YY years | | | | | |
| >=ZZ years | | | | | |
| Total | | | | | |
| Age median and range | | | | | |
| N | | | | | |
| Median (Range) | | | | | |
| Mean (std) | | | | | |
| Gender | | | | | |
| Male | | | | | |
| Female | | | | | |
| Total | | | | | |

Notes: Percentage is based on number of patients by dose level.

Table 10.2.1. 2 Supportive listing: Baseline demographics characteristic

| Dose level | Patient No. | Gender | Age at study entry (calculated) |
|------------|-------------|--------|---------------------------------|

## 10.2.2. Cancer history

Table 10.2.2. 1 Primary tumor by dose level

| | DL1 | DL2 | DL3 | | Total |
|------------------------------|------|------|------|------|-------|
| | N(%) | N(%) | N(%) | N(%) | N(%) |
| Breast cancer | | | | | |
| Epithelial ovarian cancer | | | | | |
| Head and neck | | | | | |
| NSCLC | | | | | |
| Germ cell tumors | | | | | |
| Biliary tract adenocarcinoma | | | | | |
| UKPS | | | | | |
| Cervix carcinoma | | | | | |
| GIST | | | | | |
| Urothelial cancer | | | | | |
| Total | | | | | |

Table 10.2.2. 2 Prior cancer history time differences

| | DL1 | DL2 | DL3 | • • • • • | Total |
|---|---|---|---|---|---|
| Time from diagnosis to first infusion (months) | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Mean (std) | | | | | |
| Time from last PD to first infusion (months) | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Mean (std) | | | | | |
| TTP of last prior therapy (months) | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Mean (std) | | | | | |

Table 10.2.2. 3 Other cancer history characteristics

Note: According to each tumor type.

| | DL 1 | DL2 | DL3 | • • • • • | Total |
|---------------------------|------|------|------|-----------|-------|
| | N(%) | N(%) | N(%) | N(%) | N(%) |
| Histology grade | | | | | |
| Well differentiated | | | | | |
| Moderately differentiated | | | | | |
| Total | | | | | |
| Current stage | | | | | |
| Early | | | | | |
| Locally advanced | | | | | |
| Metastatic | | | | | |
| Total | | | | | |
| TNM | | | | | |
| T1N1M1 | | | | | |
| Total | | | | | |

### 10.2.3. Sites involved

Table 10.2.3. 1 Supporting listing: Evaluation method

| | DL 1 | DL2 | DL3 | •••• | Total |
|----------------|------|------|------|------|-------|
| | N(%) | N(%) | N(%) | N(%) | N(%) |
| No. of sites | | | | | |
| 1 site | | | | | |
| 2 sites | | | | | |
| Total | | | | | |
| No. of sites | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Mean (std) | | | | | |
| Sites | | | | | |
| Lung | | | | | |
| Liver | | | | | |
| Bulky disease | | | | | |
| > 50 mm | | | | | |
| ≤50mm | | | | | |
| Total | | | | | |

Table 10.2.3. 2 Supportive listing: Sites of disease (RECIST v1.1)

| 1 autc 10.2.3. 2 | Supportiv | c fisting. Sites of disc | asc (REC | 151 VI.I) | | |
|---|---|---|---|---|---|---|
| Dose level | Patient No. | Tumor assessment date | Type* | Method | Site | Longest diameter |

<sup>(\*)</sup> Target lesion/Non target lesion.

### 10.2.4. Previous treatment summary

Table 10.2.4. 1 Previous treatment summary by dose level

| 1 uote 10.2.1. 1 11evious ite | adment summary by do | 56 16 (61 | | | |
|---|---|---|---|---|---|
| | DL1 | DL2 | DL3 | | Total |
| | N(%) | N(%) | N(%) | N(%) | N(%) |
| Systemic therapy | | | | | |
| Surgery | | | | | |
| Radiotherany | | | | | |

Notes: Percentage is based on number of patients by dose level.

Table 10.2.4. 2 Previous surgery by dose level

| | DL1 | DL2 | DL3 | | Total |
|-----|------|------|------|------|-------|
| | N(%) | N(%) | N(%) | N(%) | N(%) |
| ъ . | | | | | |

Previous surgery

Yes

No

Total

Notes: Percentage is based on number of patients by dose level.

Table 10.2.4. 3 Previous radiotherapy by dose level

| 14010 10:2: 5 110 / 10 | DI 1 | DI 2 | DI 2 | | T-4-1 |
|------------------------|------|------|------|-------------|-------|
| | DL1 | DL2 | DL3 | • • • • • • | Total |
| | N(%) | N(%) | N(%) | N(%) | N(%) |
| Previous radiotherapy | | | | | |

Yes

No Total

Notes: Percentage is based on number of patients by dose level.

Table 10.2.4. 4 Agents of previous anticancer therapies (ATC 1 & 4) by dose level

| Tuble 10. | 2. i. i rigents | Dr. 1 | DI 2 | · / · | y dose level | m · 1 | _ |
|---|---|---|---|---|---|---|---|
| | | DL 1 | DL2 | DL3 | | Total | |
| | | N(%) | N(%) | N(%) | N(%) | N(%) | _ |

ATC level 1

ATC level 2

ATC level 4

. .

ATC level 4

Notes: Percentage is based on number of patients by dose level.

Table 10.2.4. 5 No. of lines/agent of prior anticancer therapies by dose level

| | DL1 | DL2 | DL3 | | Total |
|----------------|------|------|------|------|-------|
| | N(%) | N(%) | N(%) | N(%) | N(%) |
| No. of lines | | | | | |
| 1 line | | | | | |
| 2 lines | | | | | |
| 3 lines | | | | | |
| $\geq$ 4 lines | | | | | |
| Total | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| No. of agents | | | | | |
| 0 agents | | | | | |
| 1 agent | | | | | |
| 2 agents | | | | | |
| 3 agents | | | | | |
| ≥4 agents | | | | | |
| Total | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Mean (std) | | | | | |

Notes: Percentage is based on number of patients by dose level.

# 10.2.5. Physical examination, vital signs, electrocardiogram and other tests

Table 10.2.5. 1 Physical examination by dose level

| | DL1 | DL2 | DL3 | | Total |
|---|---|---|---|---|---|
| | N(%) | N(%) | N(%) | N(%) | N(%) |
| Physical examination | | | | | |
| Normal | | | | | |
| Abnormal | | | | | |
| Total | | | | | |
| Weight (kg) | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Height (cm) | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| BSA (m <sup>2</sup> -calculated by Dubois & Dubois formula) | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| BMI | • | • | • | • | |
| N | | | | | |
| Median (range) | | | | | |
| - | • | • | • | • | • |

Notes: Percentage is based on number of patients by dose level.

Table 10.2.5. 2 ECOG performance status by dose level

| PS (ECOG) | DL1 | DL2 | DL3 | | Total |
|-----------|------|------|------|------|-------|
| PS(ECCO) | N(%) | N(%) | N(%) | N(%) | N(%) |
| 0 | | | | | |
| 1 | | | | | |
| Total | | | | | |

Notes: Percentage is based on number of patients by dose level.

Table 10.2.5. 3 Supportive listing: Patients with  $PS \ge 2$ 

| Dose level | Patient No. | Performance status (ECOG) |
|------------|-------------|---------------------------|
|------------|-------------|---------------------------|

Table 10.2.5. 4 ECG by dose level

| | DL 1 | DL2 | DL3 | | Total |
|------------------|------|------|------|------|-------|
| | N(%) | N(%) | N(%) | N(%) | N(%) |
| ECG result | | | | | |
| Abnormal | | | | | |
| Normal | | | | | |
| Total | | | | | |
| PR interval | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Mean (std) | | | | | |
| QT interval | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Mean (std) | | | | | |
| Ventricular rate | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Mean (std) | | | | | |
| QTc interval | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Mean (std) | | | | | |
Table 10.2.5. 5 LVEF by dose level

| | DL1 | DL2 | DL3 | | Total |
|----------------|------|------|------|------|-------|
| | N(%) | N(%) | N(%) | N(%) | N(%) |
| LVEF result | | | | | |
| Normal | | | | | |
| Abnormal | | | | | |
| Total | | | | | |
| LVEF method | | | | | |
| ECHO | | | | | |
| MUGA | | | | | |
| Total | | | | | |
| LVEF value | | | | | |
| N | | | | | |
| Median (range) | | | | | |
| Mean (std) | | | | | |

Table 10.2.5. 6 Vital signs by dose level

| Pulse (beats/minute): N Median (range) Mean (std) Temperature (°C): |
|-------------------------------------------------------------------------|
| Median (range)<br>Mean (std) |
| Mean (std) |
| Temperature (9C): |
| inipaddic (C). |
| N |
| Median (range) |
| Mean (std) |
| Blood pressure systolic (mmHg): |
| N |
| Median (range) |
| Mean (std) |
| Blood pressure diastolic (mmHg): |
| N |
| Median (range) |
| Mean (std) |

# 10.2.6. Hematological evaluation at baseline

Table 10.2.6. 1 Hematological abnormalities by dose level

| | | | | | DLn | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Event | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 1-2 | Grade 3-4 | Grade 1-4 | N |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | |
| Anemia | | | | | | | | | |
| Leukopenia | | | | | | | | | |
| Neutropenia | | | | | | | | | |
| Lymphopenia | | | | | | | | | |
| Thrombocytopenia | | | | | | | | | |

Table 10.2.6. 2 Median and range for hematological parameters by dose level

| Parameter | DL1 | DL2 | DL3 | <br>Total |
|----------------|-----|-----|-----|-----------|
| Hemoglobin | | | | |
| N | | | | |
| Median (range) | | | | |
| Mean (std) | | | | |
| WBC: | | | | |
| N | | | | |
| Median (range) | | | | |
| Mean (std) | | | | |
| Lymphocytes | | | | |
| N | | | | |
| Median (range) | | | | |
| Mean (std) | | | | |
| XXXXX | | | | |
| N | | | | |
| Median (range) | | | | |
| Mean (std) | | | | |

Table 10.2.6. 3 Supportive listing: Patients with grade ≥2 hematological abnormalities

| Dose level | Patient No. Lab. to | st Cycle | Examination date | Std. value | NCI-CTCAE V4.03 grade |
|---|---|---|---|---|---|

Table 10.2.6. 4 Supportive listing: Patients with missing grade for hematological abnormalities

| Dose level | Patient No. Lab. test | Cycle | Examination date | Std. value | NCI-CTCAE v4.03 grade |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

### 10.2.7. Biochemical evaluation at baseline

Table 10.2.7. 1 Biochemical abnormalities by dose level

| | | | | | DLn | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Event | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 1-2 | Grade 3-4 | Grade 1-4 | N |
| | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | N(%) | |
| AP increase | | | | | | | | | |

ALT increase AST increase

XXXXX

| Parameter | | DLI | I | )LII | DLII | I | | | | DL r | 1 | Total | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| AP | | | | | | | | | | | | | |
| N | | | | | | | | | | | | | |
| Median (range) | | | | | | | | | | | | | |
| Mean (std) | | | | | | | | | | | | | |
| ALT | | | | | | | | | | | | | |
| N | | | | | | | | | | | | | |
| Median (range) | | | | | | | | | | | | | |
| Mean (std) | | | | | | | | | | | | | |
| AST | | | | | | | | | | | | | |
| N<br>Madian ( | | | | | | | | | | | | | |
| Median (range) | | | | | | | | | | | | | |
| Mean (std) XXXXXXXX | | | | | | | | | | | | | |
| naaaaa<br>N | | | | | | | | | | | | | |
| Median (range) | | | | | | | | | | | | | |
| Mean (std) | | | | | | | | | | | | | |
| • | | | | | | | | | | | | | |
| Table 10.2.7. | 3 Support | ive listi | ng· Pati | ients | with grade | e >2 bioc | chemic | al ahn | ormal | ities | | | |
| | ** | | | | | | | | | | CI-CT0 | CAE | V4.0 |
| Dose level | Patient No. | Lab. test | : C | ycle | Examination | n date | Std. v | alue | xULN | | ade | C7 IL | V 1.0 |
| Table 10.2.7. | 4 Support | ive listi | ng: Pati | ients | with miss | ing grade | e for b | iochen | nical a | | | | 374.0 |
| | 4 Support Patient No. | | | ients<br>Ycle | | ing grade | | iochen<br>Std. va | | N | nalitie:<br>CI-CTO<br>ade | | V4.0 |
| | | | | | | | | | | N | CI-CT0 | | V4.0 |
| Dose level | | Lab. test | C | Ycle | Exan | | | | | N | CI-CT0 | | V4.0 |
| Dose level | Patient No. 8. Signs a | Lab. test | : C | Sycle | Exan | | | | | N | CI-CT0 | | V4.0 |
| 10.2.3 Table 10.2.8. MedDRA System | Patient No. 8. Signs a | nd sym | : C | s at | Exan | | | | | N<br>gr | CI-CT0 | | |
| 10.2.3 Table 10.2.8. MedDRA Systen | Patient No. 8. Signs a | nd sym | nptoms | s at | Exan baseline se level | nination da | | Std. va | ilue | N<br>gr | CI-CTO<br>ade | CAE | |
| 10.2.3 Table 10.2.8. MedDRA Systen | Patient No. 8. Signs a | nd sym | nptoms | s at | Exan baseline se level DL II | nination dat | | Std. va | ilue | N<br>gr<br>DI | CI-CTO<br>ade | Tota | ıl |
| 10.2.3 Table 10.2.8. MedDRA Systen | Patient No. 8. Signs a | nd sym | nptoms | s at | Exan baseline se level DL II | nination dat | | Std. va | ilue | N<br>gr<br>DI | CI-CTO<br>ade | Tota | ıl |
| 10.2.3 Table 10.2.8. MedDRA Systen | Patient No. 8. Signs a | nd sym | nptoms | s at | Exan baseline se level DL II | nination dat | | Std. va | ilue | N<br>gr<br>DI | CI-CTO<br>ade | Tota | ıl |
| 10.2.s Table 10.2.8. MedDRA System Preferred Term | Patient No. 8. Signs a 1 Signs ar n Organ Class | nd sym | nptoms<br>otoms b | s at y do: " " | Exan baseline se level DL II N % | nination dat | | Std. va | ilue | N<br>gr<br>DI | CI-CTO<br>ade | Tota | ıl |
| 10.2.s Table 10.2.8. MedDRA System Preferred Term | Patient No. 8. Signs a 1 Signs ar n Organ Class | nd sym | nptoms<br>otoms b | s at y do: " " | Exan baseline se level DL II N % | nination dat | | Std. va | ilue | N<br>gr<br>DI | CI-CTO<br>ade | Tota | ıl |
| 10.2.s Table 10.2.8. MedDRA System Preferred Term | Patient No. 8. Signs a 1 Signs ar n Organ Class | nd sym | nptoms<br>otoms b | s at y do: " " | Exan baseline se level DL II N % | nination dat | | Std. va | ilue | N<br>gr<br>DI | CI-CTO<br>ade | Tota | ો |
| 10.2.s<br>Table 10.2.8.<br>MedDRA System<br>Preferred Term | Patient No. 8. Signs a 1 Signs ar n Organ Class | nd sym | nptoms<br>otoms b | s at y do: " " | Exan baseline se level DL II N % | nination dat | | Std. va | ilue | N<br>gr<br>DI | CI-CTO<br>ade | Tota | ો |
| 10.2.8 Table 10.2.8. MedDRA System Preferred Term | Patient No. 8. Signs at Signs arn Organ Classes et is based on nu | nd sym | nptoms otoms b DL1 N | s at y do: y dose | Exan baseline se level DL II N % | DL III | N | Std. va | <br>N % | N<br>gr<br>DI | CI-CTO<br>ade | Tota | ો |
| Table 10.2.7. 4 Dose level 10.2.8 Table 10.2.8. MedDRA System Preferred Term Notes: Percentage | Patient No. 8. Signs at Signs at Organ Class e is based on nu. | nd sympole of grade | nptoms otoms b DL1 N | s at y do: | baseline se level DL II N % | DL III | ns and | % Std. va | <br>N % | DI<br>6 N | L n | Tota<br>N | ત્રી % |
| 10.2.8 Table 10.2.8. MedDRA System Preferred Term | Patient No. 8. Signs at Signs arn Organ Classes et is based on nu | nd sympole of grade | nptoms otoms b DL1 N | s at y dose y dose A not | baseline se level DL II N % | DLIII N % | <br>N | % Std. va | <br>N % | N<br>gr<br>DI | L n | Tota | 9/0 |

| Dose level | Patient No. | Literal | MedDRA<br>Preferred Term | NCI-CTCAE<br>V4.03<br>grade | Start date | Disease-related |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

Table 10.2.8. 3 Incidence of signs and symptoms by dose level

| MedDRA | Syste | emDL | Ι | | | | | | - | | | | | | | | | DL | n | | | | | | | Tot | tal | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Organ Class | - | Gr. | 1 | Gr. | 2 | Gr. | 3 | Gr. | 4 | Gr. | 1 | Gr. | 2 | Gr. | 3 | Gr. | 4 | Gr. | 1 | Gr. | 2 | Gr | 3 | Gr. | 4 | Gr. | 1 | Gr. | 2 | Gr. | 3 | Gr. 4 | Į. |
| Preferred Tem | n | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |

Notes: Percentage is based on number of patients by dose level.

### 10.2.9. Concomitant medication starting pre-study

Table 10.2.9. 1 Concomitant medication starting pre-study (ATC 1 and 4) by dose level

| Medication Term | Medication Term | Medication Term | DLI | | DLII | | DLIII | | | | | | DL n | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (ATC level 1) | (ATC level 2) | (ATC level 4) | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

Notes: Percentage is based on number of patients by dose level.

Table 10.2.9. 2 Concomitant medication starting pre-study (Transfusions and/or EPO)

| Medication Term | Medication Term | Medication Term | DLI | | DLII | | DLIII | | | | | | DL n | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (ATC level 1) | (ATC level 2) | (ATC level 4) | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

Platelet transfusion

RBC transfusion

EPO

Notes: Percentage is based on number of patients by dose level

Table 10.2.9. 3 Supportive listing: Patients with transfusions and/or EPO (pre-study)

| Dose level | Patient No. | Cycle | Туре | Literal term | ATC 4 | ATC2 | ATC 1 | Route | Dose | Unit | Start date | End date | Reason for use |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

## 11. APPENDIX II. SAFETY EVALUATION

## 11.1. Extent of exposure

### 11.1.1. Cumulative Dose, Dose Intensity and Relative Dose Intensity: PM060184

Table 11.1.1. 1 No. of cycles administered (PM060184)

| | | Patients | Cycles |
|---|---|---|---|
| Dose level | No. of cycles infused | No. of patients No. of patients (accumulated) | No. of cycles No. of cycles (accumulated) |
| I | 1 cycle | | |
| | 2 cycles | | |
| II | 1 cycle | | |
| | 2 cycles | | |
| III | 1 cycle | | |
| | 2 cycles | | |
| N | 1 cycle | | |
| | 2 cycles | | |
| Total | 1 cycle | | |
| | 2 cycles | | |
| | 3 cycles | | |
| | N cycles | | |

Table 11.1.1. 2 No. of cycles administered by dose level (PM060184)

| No. | of cyclesDL I | | DLI | I | 1 11 1 | II | | | | | DL: | n | Total | ĺ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| administer | ed per patient N | % | N | % | N | % | N | % | N | % | N | % | N | % |
| 1 ovele | | | | | | | | | | | | | | |

1 cycle

2 cycles

3 cycles

N cycles

N

Median (range)

Mean (std)

Notes: Percentage is based on number of patients by dose level.

Table 11.1.1.3 Cumulative dose, DI and RDI by dose level (PM060184)

| Table 11.1.1. 5 Cumulan | ive dose, D | i aliu KDi ( | by dosc icvi | JI (I IVIOOO | 104) | | |
|---|---|---|---|---|---|---|---|
| | DLI | DLII | DLIII | | | DL n | Total |
| Cumulative dose (mg/m²) | | | | | | | |
| N | | | | | | | |
| Median (range) | | | | | | | |
| Mean (std) | | | | | | | |
| Dose intensity (mg/m²/week) | | | | | | | _ |
| N | | | | | | | |
| Median (range) | | | | | | | |
| Mean (std) | | | | | | | |
| Relative dose intensity (%) | | | | | | | _ |
| N | | | | | | | |
| Median (range) | | | | | | | |
| Mean (std) | | | | | | | |

| Table 11 1 1 4 | Supportive listing: | Patients with less | than 60% of RI | OL (PM060184) |
|---|---|---|---|---|
| 1 aut 11.1.1.4 | Supportive fishing. | Tauchts with 1055 | man ou /o oi Ki | )1 (1 WIUUU10 <del>4</del> ) |

| | | Intended doce | Total | Delay/OmissionDose | Dose |
|---|---|---|---|---|---|
| Dose level Patient No. | Cycle | Date Intended dose | dose | Delay/Omission : | modification |
| | | (mg/m²) | (mg) | specify modification | specify |

## 11.1.2. Cumulative Dose, Dose Intensity and Relative Dose Intensity: Gemcitabine

Table 11.1.2. 1 No. of cycles administered (gemcitabine)

| | | Patients | Cycles |
|---|---|---|---|
| Dose level | No. of cycles infused | No. of patients No. of patients (accumulated) | No. of cycles No. of cycles (accumulated) |
| I | 1 cycle | | |
| | 2 cycles | | |
| II | 1 cycle | | |
| | 2 cycles | | |
| III | 1 cycle | | |
| | 2 cycles | | |
| N | 1 cycle | | |
| | 2 cycles | | |
| Total | 1 cycle | | |
| | 2 cycles | | |
| | 3 cycles | | |
| | N cycles | | |

| No. | of | cyclesDL1 | | DL. | 1 | DLI | Ш | | | • • • • | | DL 1 | n | Lota | l |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| admini | stered p | er patient N | % | N | % | N | % | N | % | N | % | N | % | N | % |
| 1 cycle<br>2 cycle<br>3 cycle | ; | | | | | | | | | | | | | | |
| 2 cycle | S | | | | | | | | | | | | | | |
| 3 cycle | S | | | | | | | | | | | | | | |
| N cycle | es | | | | | | | | | | | | | | |

N

Median (range)

Mean (std)

Table 11.1.2. 3 Cumulative dose, DI and RDI by dose level (gemcitabine)

| | DLI | DLII | DLIII | <br> | DL n | Total |
|-----------------------------|-----|------|-------|------|------|-------|
| Cumulative dose (mg/m²) | | | | | | |
| N | | | | | | |
| Median (range) | | | | | | |
| Mean (std) | | | | | | |
| Dose intensity (mg/m²/week) | | | | | | |
| N | | | | | | |
| Median (range) | | | | | | |
| Mean (std) | | | | | | |
| Relative dose intensity (%) | | | | | | |
| N | | | | | | |
| Median (range) | | | | | | |
| Mean (std) | | | | | | |

Table 11.1.2. 4 Supportive listing: Patients with less than 60% of RDI (gemcitabine)

| Dose level Patient No. | Cycle | Date | Intended dose<br>(mg/m²) | Total dose<br>(mg) Delay | Delay<br>specify | Dose<br>modification | Dose<br>modification<br>specify |
|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|

### 11.1.3. Cycle Delays: PM060184

Note: "Dose Delayed: No/Yes" in the CRF will be used to calculate the delay. For cycles considered as delayed by the Investigator, the delay will be calculated as:

Delay = (Date of current drug administration) - (Date of previous drug administration) - theoretical cycle duration in days (21))

A second internal analysis taking into account the drug administration dates rather than the item "dose delay" completed by the Investigator will be performed in order to know the real delay occurred, in days.

Note: The distribution of delays according to the administered cycle will be studied by means of counts and percentages. The reason for cycle delay will be detailed, specifying how many delays were due to treatment and how many were not. Within delays attributable to the study drug, hematological and non-hematological reasons will be outlined and the exact reason will be stated (specific data listings will be provided).

| Table 11.1.3. 1 | Summary of dose dela | y by dose level | (PM060184) |
|-----------------|----------------------|-----------------|------------|
| Dose delay | DL1 | DLII | DLIII |

No. of patients

No. of patients susceptible to be delayed

No. of patients with delay (n,%)

- => Hematological tox (n,%)
- > Non-hematological tox (n,%)
- =>Both (n,%)
- > Non drug-related (n,%)

Patients with 1 cycle delayed (n,%)

Patients with 2 cycles delayed (n,%)

Patients with 3 cycles delayed (n,%)

Patients with 4 cycles delayed (n,%) Summary statistics no. of cycles delayed

No. of cycles

No. of cycles susceptible to be delayed

No. of cycles with delay (n,%)

- => Hematological tox (n,%)
- > Non-hematological tox (n,%)
- => Both (n,%)
- $\Longrightarrow$  Non drug-related (n,%)

Notes: Percentage is based on number of patients by dose level.

- \* Drug-related.
- \*\* Non drug-related.

Table 11.1.3. 2 Supportive listing: Dose delays (PM060184)

| Dose level | Patient No. | Cycle/Day | Date | Intended dose<br>(mg/m²) | Total dose (mg) | Length of delay | Delay<br>reason | Delay specify |
|---|---|---|---|---|---|---|---|---|

. . .

Total

Table 11.1.3. 3 Supportive listing: Dose delays excluding administrative reasons (PM060184)

| Dogo lovol | Dationt No. | Cyala/Day | Doto | Intended dose | Total dose | Length of | Delay | Delay specify |
|---|---|---|---|---|---|---|---|---|
| Dose level | Pauent No. | Cycle/Day | Date | $(mg/m^2)$ | (mg) | delay | reason | Delay specify |

<sup>(\*)</sup> Excluding administrative reasons.

11.1.4.

# **Cycle Delays: Gemcitabine**

Table 11.1.4. 1 Summary of dose delay by dose level (gemcitabine)

| Dose delay | DLI | DLII | DLIII | <br>Total |
|---|---|---|---|---|
| No. of patients | DLI | DEII | DLIII | Tout |
| No. of patients susceptible to be delayed | | | | |
| No. of patients with delay (n,%) | | | | |
| => Hematological tox (n,%) | | | | |
| => Non-hematological tox (n,%) | | | | |
| => Both (n,%) | | | | |
| => Non drug-related (n,%) | | | | |
| Patients with 1 cycle delayed (n,%) | | | | |
| Patients with 2 cycles delayed (n,%) | | | | |
| Patients with 3 cycles delayed (n,%) | | | | |
| Patients with 4 cycles delayed (n,%) | | | | |
| Summary statistics no. of cycles delayed | | | | |
| No. of cycles | | | | |
| No. of cycles susceptible to be delayed | | | | |
| No. of cycles with delay (n,%) | | | | |
| $\Longrightarrow$ Hematological tox (n,%) | | | | |
| $\Longrightarrow$ Non-hematological tox (n,%) | | | | |
| ⇒> Both (n,%) | | | | |
| > Non drug-related (n,%) | | | | |
| Notes: Percentage is based on number of pa | atients by dose | level. | | |

Table 11.1.4. 2 Supportive listing: Dose delays (gemcitabine)

| Dose level Patient No. | Cycle/Day Date | Intended dose<br>(mg/m²) | Total dose<br>(mg/m²) | Length of delay | Delay<br>reason | Delay specify |
|---|---|---|---|---|---|---|

Table 11.1.4. 3 Supportive listing: Dose delays excluding administrative reasons (gemcitabine)

| Dose level Patient No. | Cycle/Day Date | Intended dose | Total dose | Length of | Delay | Dolov morify |
|---|---|---|---|---|---|---|
| Dose level Patient No. | Cycle/Day Date | $(mg/m^2)$ | $(mg/m^2)$ | delay | reason | Delay specify |

<sup>(\*)</sup> Excluding administrative reasons.

<sup>\*</sup> Drug-related.
\*\* Non drug-related.

## 11.1.5. Dose Omission: PM060184

Table 11.1.5.1. Summary of dose omission by dose level (PM060184).

| Dose omission | DLI | DLII | DLIII | <br>Total |
|-------------------------------------------|-----|------|-------|-----------|
| No. of patients | | | | |
| No. of patients susceptible to be omitted | | | | |
| No. of patients with omission (n,%) | | | | |
| => Hematological tox (n,%) | | | | |
| > Non-hematological tox (n,%) | | | | |
| ⇒Both (n,%) | | | | |
| > Non drug-related (n,%) | | | | |
| Patients with 1 cycle omitted (n,%) | | | | |
| Patients with 2 cycles omitted (n,%) | | | | |
| Summary statistics no. of cycles omitted | | | | |
| No. of cycles | | | | |
| No. of cycles susceptible to be omitted | | | | |
| No. of cycles with omission (n,%) | | | | |
| => Hematological tox (n,%) | | | | |
| > Non-hematological tox (n,%) | | | | |
| ⇒> Both (n,%) | | | | |
| >> Non drug-related (n,%) | | | | |

Notes: Percentage is based on number of patients by dose level.

Table 11.1.5. 2 Listing of dose omissions (PM060184)

<sup>\*</sup> Drug-related.
\*\* Non drug-related.

### 11.1.6. Dose Omission: Gemcitabine

Table 11.1.6. 1 Summary of dose omission by dose level (gemcitabine)

| Dose omission | DLI | DLII | DLIII | | Total |
|---|---|---|---|---|---|
| No. of patients | | | | | |
| No. of patients susceptible to be omitted | | | | | |
| No. of patients with omission $(n,\%)$ | | | | | |
| =>Hematological tox (n,%) | | | | | |
| => Non-hematological tox (n,%) | | | | | |
| =>Both (n,%) | | | | | |
| => Non drug-related (n,%) | | | | | |
| Patients with 1 cycle omitted (n,%) | | | | | |
| Patients with 2 cycles omitted (n,%) | | | | | |
| Summary statistics no. of cycles omitted | | | | | |
| No. of cycles | | | | | |
| No. of cycles susceptible to be omitted | | | | | |
| No. of cycles with omission $(n,\%)$ | | | | | |
| =>Hematological tox | | | | | |
| => Non-hematological tox (n,%) | | | | | |
| $\Longrightarrow$ Both (n,%) | | | | | |
| => Non drug-related (n,%) | | | | | |
| Notes: Percentage is based on number of nations | by doce level | | | • | |

Notes: Percentage is based on number of patients by dose level.

Table 11.1.6. 2 Listing of dose omissions (gemcitabine)

| Table 11.1.6. 2 | Listing of do | se omissions (ge | emcitabine) | | |
|---|---|---|---|---|---|
| Dose level | Patient No. | Cycle/Day | Infusion No | Reason for omission | Specify |

<sup>\*</sup> Drug-related.

<sup>\*\*</sup> Non drug-related.

#### 11.1.7. Dose Modification: PM060184

All dose modifications will be considered and described, specifying the reason for change (hematological toxicity, non-hematological toxicity or other causes not due to the study drug) and the exact reason will be stated (specific data listings will be provided).

Table 11.1.7. 1 Summary of reduced cycles by dose level (PM060184)

| Dose reduction | DLI | DLII | DLIII | <br>Total |
|-------------------------------------------|-----|------|-------|-----------|
| No. of patients | | | | |
| No. of patients susceptible to be reduced | | | | |
| No. of patients with reduction (n,%) | | | | |
| =>Hematological tox (n,%) | | | | |
| > Non-hematological tox (n,%) | | | | |
| ⇒Both (n,%) | | | | |
| $\Longrightarrow$ Non drug-related (n,%) | | | | |
| Patients with 1 cycle reduced (n,%) | | | | |
| Patients with 2 cycles reduced (n,%) | | | | |
| Summary statistics no. of cycles reduced | | | | |
| No. of cycles | | | | |
| No. of cycles susceptible to be reduced | | | | |
| No. of cycles with reduction (n,%) | | | | |
| =>Hematological tox (n,%) | | | | |
| > Non-hematological tox (n,%) | | | | |
| ⇒Both (n,%) | | | | |
| > Non drug-related (n,%) | | | | |

Table 11.1.7. 2 Listing of dose reductions (PM060184)

| Dose level | Patient No. | Cycle/Day | Start date | Is infusion reduced? | Reduce reason | Specify |
|---|---|---|---|---|---|---|

#### 11.1.8. Dose Modification: Gemcitabine

All dose modifications will be considered and described, specifying the reason for change (hematological toxicity, non-hematological toxicity or other causes not due to the study drug) and the exact reason will be stated (specific data listings will be provided).

Table 11.1.8. 1 Summary of reduced cycles by dose level (gemcitabine)

| Dose reduction | DLI | DLII | DLIII | <br>Total |
|---|---|---|---|---|
| No. of patients | | | | |
| No. of patients susceptible to be reduced | | | | |
| No. of patients with reduction (n,%) | | | | |
| ==> Hematological tox (n,%) | | | | |
| > Non-hematological tox (n,%) | | | | |
| ⇒Both (n,%) | | | | |
| > Non drug-related (n,%) | | | | |
| Patients with 1 cycle reduced (n,%) | | | | |
| Patients with 2 cycles reduced (n,%) | | | | |
| Summary statistics no. of cycles reduced | | | | |
| No. of cycles | | | | |
| No. of cycles susceptible to be reduced | | | | |
| No. of cycles with reduction (n,%) | | | | |
| ==>Hematological tox (n,%) | | | | |
| $\Longrightarrow$ Non-hematological tox (n,%) | | | | |
| ⇒Both (n,%) | | | | |
| > Non drug-related (n,%) | | | | |

Table 11.1.8. 2 Listing of dose reductions (gemcitabine)

| Dose level | Patient No. | Cycle/Day | Start date | Is infusion reduced? | Reduce reason | Specify |
|---|---|---|---|---|---|---|

# 11.2. Dose-limiting toxicities (DLT)

# 11.2.1. Dose-limiting toxicities

Table 11.2.1. 1 Summary of patients with DLT by dose level

| Dose level | | Escalation fa | ctor | N | DLT |
|---|---|---|---|---|---|
| Note: Each row show | vs the number of patients o | f that dose level, the nu | umber of cases with defined DL | Ts of the N | patients. |
| T. 1. 1. 2. 2 | D . I . CDI.T | | | | |
| Table 11.2.1. 2 | Details of DLT | | | | |
| | | DLT description | NCI-CTCAE V4.03 grade | | |

## 11.3. Adverse events (AEs)

## 11.3.1. Display of adverse events

Table 11.3.1. 1 Drug-related (or relationship UK) AEs. Worst grade by patient

| MadDDA Castone Oregon Class | DLI | | | | | | | | DLn | | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class | Gr. 1 | Gr.2 | Gr.3 | Gr.4 | Gr. 1 | Gr.2 | Gr.3 | Gr.4 | Gr. 1 | Gr.2 ( | Gr. 3 Gr. 4 | Gr. 1 | Gr.2 | Gr.3 | Gr.4 |
| Preferred Term | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % r | n % n | % n % | n % | n % | n % |

Table 11.3.1.2 Drug-related (or relationship UK) AEs in the first cycle

| MedDRA System Organ Class | DLI | | | | | | | | DLn | | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | Gr. 1 | Gr.2 | Gr. 3 | Gr.4 | Gr. 1 | Gr.2 | Gr. 3 | Gr. 4 | Gr. 1 | Gr.2 | Gr. 3 Gr. 4 | Gr. 1 | Gr.2 | Gr.3 | Gr.4 |
| Ficiality Italii | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % n | n % n % | 6 n % | n % | n % | n % |

Table 11.3.1. 3 Drug-related (or relationship UK) AEs. Worst grade per cycle

| MedDRA System Organ Class | DLI | | | | | | | | DLn | | To | tal | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | Gr. 1 | Gr. 2 | Gr. 3 | Gr.4 | Gr. 1 | Gr.2 | Gr. 3 | Gr.4 | Gr. 1 | Gr. 2 Gr. 3 | Gr.4 Gr | .1 Gr.2 | Gr.3 | Gr.4 |
| Fieldied Telli | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % n % | 6 n % n | % n % | n % | n % |

| Table 11.3.1. 4 | Drug related | (or relationship | pUK) | AEs in $\geq 10\%$ of p | atients |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

| MadDDA Stratova Ownor Class | DLI | | | | | | | | DLn | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class<br>Preferred Term | Gr. 1 | Gr. 2 | Gr.3 | Gr.4 | Gr. 1 | Gr.2 | Gr. 3 | Gr.4 | Gr. 1 | Gr.2 Gr.: | 3 Gr. 4 | Gr. 1 Gr. 2 | Gr.3 | Gr.4 |
| Hadia falli | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % n | % n % | n % n % | n % | n % |

Notes: Percentage is based on number of patients by dose level.

Table 11.3.1. 5 Drug related (or relationship UK) AEs in ≥10% of patients. Worst grade per cycle

| MadDD A Contacta Orecon Class | DLI | | | | | | | | DLn | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class<br>Preferred Term | Gr. 1 | Gr. 2 | Gr. 3 | ìr.4 | Gr. 1 | Gr.2 | Gr.3 | Gr.4 | Gr. 1 | Gr. 2 | Gr. 3 Gr. 4 | Gr. 1 Gr. 2 | Gr. 3 | Gr.4 |
| Ficiality Telli | n % | n % | n % n | 1 % | n % | n % | n % | n % | n % | n % | n % n % | % n % n % | n % | n % |

Notes: Percentage is based on number of cycles by dose level.

Table 11.3.1. 6 AEs regardless of relationship. Worst grade by patient

| MadDDA Costone Overen Class | DLI | | | | | | | | DLn | | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class<br>Preferred Term | Gr. 1 | Gr. 2 | Gr. 3 | Gr.4 | Gr. 1 | Gr.2 | Gr. 3 | Gr. 4 | Gr. 1 | Gr.2 | Gr. 3 Gr. 4 | Gr. 1 | Gr.2 | Gr.3 | Gr.4 |
| Ficiality Talli | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % n | % n % | n % | n % | n % |

| MedDRA System Organ Class | DLI | | | | | | | | DLn | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | Gr. 1 | Gr. 2 | Gr.3 | Gr.4 | Gr. 1 | Gr.2 | Gr. 3 | Gr.4 | Gr. 1 | Gr.2 Gr. | .3 Gr.4 | Gr. 1 Gr. 2 | Gr.3 | Gr.4 |
| Ticicia Taili | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % n | % n % | n % n % | n % | n % |

Notes: Percentage is based on number of patients by dose level.

Table 11.3.1. 8 AEs regardless of relationship. Worst grade per cycle

| M IDDA DI I | | | | | | | | DI | | | | Tr 4 1 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA DLI | | | | | | | | DLn | | | | Total | | | |
| System Organ <sub>Gr. 1</sub> | Gr.2 | Gr. 3 | Gr.4 | Gr. 1 | Gr. 2 | Gr. 3 | Gr.4 | Gr. 1 | Gr.2 | Gr. 3 | Gr.4 | Gr. 1 | Gr. 2 | Gr 3 | Gr.4 |
| Class | O | 01.0 | O | O1. 1 | O | 01.0 | | | | | | | O <b>-</b> | 01.0 | O |
| Preferred Term n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % |

Notes: Percentage is based on number of cycles by dose level.

Table 11.3.1. 9 AEs observed in ≥10% of cycles

| MadDD A Contain Organ Class | DLI | | | | | | | | DLn | | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class<br>Preferred Term | Gr. 1 | Gr.2 | Gr.3 | Gr.4 | Gr. 1 | Gr.2 | Gr.3 | Gr. 4 | Gr. 1 | Gr.2 | Gr. 3 | Gr.4 | Gr. 1 Gr. 2 | Gr.3 | Gr.4 |
| ricialati falli | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % n % | n % | n % |

Notes: Percentage is based on number of cycles by dose level. Table 11.3.1. 11 Supportive listing: Drug-related (or relationship UK) grade 2-4 AEs MedDRA NCI-CTCAE SAE Relationship to Main Preferred Term Literal term Patient No. Cycle Dose level SOC Onset date Resolved date Action taken V4.03 grade study drug (Y/N) consequence

NCI-CTCAE SAE

(Y/N)

V4.03 grade

Gr. 1

Literal term

Gr.4

Gr. 3

MedDRA

Preferred Term

Gr. 2

Gr.3

Gr. 4

DLn

Gr. 1

Gr.2

Gr. 3

Resolved date

Onset date

Gr.4

Total

Gr. 1

Relationship to

study drug

Gr.2

Gr.3

Main

consequence

Action taken

Gr. 4

Table 11.3.1. 10 AEs observed in ≥10% of patients. Worst grade per cycle

Table 11.3.1. 12 Supportive listing: All AEs regardless of relationship

Cycle

SOC

MedDRA System Organ Class

Preferred Term

Dose level

Patient No.

DLI

Gr. 1

## 11.4. Deaths and other serious adverse events

## 11.4.1. Deaths

| Oose level Patient No. | Last cycle received | Last infusion date | Death date | Time from last infusion date (days) | Cause | Comments | Time on study (weeks) |
|---|---|---|---|---|---|---|---|
| ote: Patient with Death rep | orted as End of Treat | ment Reason. | | | | | |
| _ | | | | | | | |
| able 11.4.1. 2 Patie | ents who died wi | thin 30 days of last dr | rug administrati | on | | | |
| | Lastavala | Last infusion | | Time from last infusion | | | |
| ose level Patient No. | Last cycle received | date | Death date | date (days) | Cause | Comments | Time on study (weeks) |
| Pose level Patient No. | - | | Death date | | Cause | Comments | Time on study (weeks) |
| Pose level Patient No. | - | | Death date | | Cause | Comments | Time on study (weeks) |
| Dose level Patient No. | - | | Death date | | Cause | Comments | Time on study (weeks) |
| | received | | Death date | | Cause | Comments | Time on study (weeks) |
| Гаble 11.4.1. 3 Listi | - | date | Death date | | Cause | Comments Time on study | Time on study (weeks) Time from last infusion |

### 11.4.2. Serious adverse events

Table 11.4.2. 1 Drug-related (or relationship UK) SAEs. Worst grade by patient

| MedDRA System Organ Class | DLI | | | | | | | | DLn | | Tot | al | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <i>y</i> | Gr. 1 | Gr. 2 | Gr.3 | Gr.4 | Gr. 1 | Gr.2 | Gr. 3 | Gr.4 | Gr. 1 | Gr.2 Gr.3 | Gr.4 Gr. | 1 Gr. 2 | Gr.3 | Gr.4 |
| Preferred Term | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % n % | % n % n | % n % | n % | n % |

Table 11.4.2. 2 Drug-related (or relationship UK) SAEs in the first cycle

| MedDRA System Organ Class | DLI | | | | | | | | DLn | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | Gr. 1 | Gr. 2 | Gr.3 | Gr.4 | Gr. 1 | Gr.2 | Gr. 3 | Gr. 4 | Gr. 1 | Gr.2 | Gr. 3 Gr. 4 | Gr. 1 G | Gr. 2 Gr. 3 | Gr.4 |
| Ficiality faili | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % n | % n % | 6 n % n | % n % | n % |

Table 11.4.2. 3 Drug-related (or relationship UK) SAEs. Worst grade per cycle

| MedDRA System Organ Class | DLI | | | | | | | | DLn | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | Gr. 1 | Gr.2 | Gr.3 | Gr.4 | Gr. 1 | Gr.2 | Gr. 3 | Gr.4 | Gr. 1 | Gr.2 Gr. | .3 Gr.4 | Gr. 1 Gr. 2 | Gr. 3 | Gr.4 |
| Hadiai Talli | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % n | % n % | 6 n % n | % n % | n % |

| Table 11.4.2. 4 | Drug related ( | or relationship Ul | K) SAEs in $\geq 10\%$ of | patients |
|---|---|---|---|---|
|---|---|---|---|---|

| ModDD A System Owen Class | DLI | | | | | | | | DLn | | | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class<br>Preferred Term | Gr. 1 | Gr.2 | Gr.3 | Gr.4 | Gr. 1 | Gr.2 | Gr. 3 | Gr. 4 | Gr. 1 | Gr.2 | Gr. 3 | Gr.4 | Gr. 1 | Gr.2 | Gr.3 | Gr.4 |
| Hada falli | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % |

Notes: Percentage is based on number of patients by dose level.

Table 11.4.2. 5 Drug related (or relationship UK) SAEs in ≥10% of patients. Worst grade per cycle

| MadDD A Crateria Overen Class | DLI | | | | | | | | DLn | | | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class<br>Preferred Term | Gr. 1 | Gr.2 | Gr.3 | Gr. 4 | Gr. 1 | Gr.2 | Gr. 3 | Gr.4 | Gr. 1 | Gr.2 | Gr.3 | Gr.4 | Gr. 1 | Gr. 2 | Gr. 3 | Gr. 4 |
| Hadia Talli | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % |

Notes: Percentage is based on number of cycles by dose level.

Table 11.4.2. 6 SAEs regardless of relationship. Worst grade by patient

| MadDDA Chartages Ourses Class | DLI | | | | | | | | DLn | | | - | <b>Fotal</b> | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class<br>Preferred Term | Gr. 1 ( | Gr. 2 | Gr.3 | Gr.4 | Gr. 1 | Gr.2 | Gr. 3 | Gr. 4 | Gr. 1 | Gr.2 | Gr. 3 | Gr. 4 ( | Gr. 1 Gr. 2 | Gr.3 | Gr.4 |
| Tieldica Tailli | n % r | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % n | ı % ı | n % n % | 6 n % | n % |

| MadDDA Castern Organ Class | DLI | | | | | | | | DLn | | | | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class<br>Preferred Term | Gr. 1 | Gr. 2 | Gr.3 | Gr.4 | Gr. 1 | Gr.2 | Gr. 3 | Gr. 4 | Gr. 1 | Gr.2 | Gr.3 | Gr. 4 | Gr. 1 Gr. 2 | Gr.3 | Gr.4 |
| Ficiality Talli | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % n % | 6 n % | n % |

Notes: Percentage is based on number of patients by dose level.

Table 11.4.2. 8 SAEs regardless of relationship. Worst grade per cycle

| MedDRA DLI | | | • | | * | | | DLn | | | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System OrganGr. 1 | Gr. 2 | Gr. 3 | Gr.4 | Gr. 1 | Gr. 2 | Gr. 3 | Gr.4 | Gr. 1 | Gr. 2 | Gr. 3 | Gr.4 | Gr. 1 | Gr. 2 | Gr.3 | Gr.4 |
| Class<br>Preferred Term <sup>n</sup> % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % |

Notes: Percentage is based on number of cycles by dose level.

Table 11.4.2. 9 SAEs observed in ≥10% of cycles

| MadDDA Contact Orecon Class | DLI | | | | | | | | DLn | | | Total | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System Organ Class<br>Preferred Term | Gr. 1 | Gr.2 | Gr. 3 | Gr. 4 | Gr. 1 | Gr.2 | Gr. 3 | Gr. 4 | Gr. 1 | Gr.2 | Gr. 3 Gr. 4 | Gr. 1 | Gr.2 | Gr.3 | Gr.4 |
| FICIGION FOILI | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % 1 | n % n % | 6 n % | n % | n % | n % |

Table 11.4.2. 10 SAEs observed in ≥10% of patients. Worst grade per cycle

| MedDRA System Organ Class | DLI | - | | | | | | | DLn | | Tota | al | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | Gr. 1 | Gr.2 | Gr. 3 | Gr. 4 | Gr. 1 | Gr. 2 | Gr.3 | Gr.4 | Gr. 1 | Gr. 2 Gr. 3 | Gr. 4 Gr. | 1 Gr. 2 | Gr.3 | Gr.4 |
| Hadiai falli | n % | n % | n % | n % | n % | n % | n % | n % | n % | n % n % | 6 n % n | % n % | n % | n % |

Notes: Percentage is based on number of cycles by dose level.

Table 11.4.2. 11 All SAEs

| | MedDRA System | | NCI- | | | | | |
|---|---|---|---|---|---|---|---|---|
| Dose level Patient No. Cycle | Organ Class | Preferred Term | CTCAE AE Status | AE relationship | AE consequences | SAE | Onset date | Resolved date |
| | OlganClass | | V4.03 grade | | | | | |

## 11.5. Clinical laboratory evaluation

### 11.5.1. Hematological abnormalities

Table 11.5.1. 1 Hematological abnormalities: Worst grade per patient

| | DLn | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Event | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 1-2 | Grade 3-4 | Grade 1-4 | N |
| Anemia | | | | | | | | | |
| Leukopenia | | | | | | | | | |
| Neutropenia | | | | | | | | | |
| Lymphopenia | | | | | | | | | |
| XXXXX | | | | | | | | | |

Notes: Percentage is based on number of patients by dose level.

Table 11.5.1. 2 Hematological abnormalities: Worst grade per cycle

| | DLn | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Event | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 1-2 | Grade 3-4 | Grade 1-4 | N |
| Anemia | | | | | | | | | |
| Leukopenia | | | | | | | | | |
| Neutropenia | | | | | | | | | |
| Lymphopenia | | | | | | | | | |
| XXXXX | | | | | | | | | |

Notes: Percentage is based on number of patients by dose level.

Table 11.5.1. 3 Supportive listing: Patients with grade ≥3 hematological abnormalities

| Dose level | Patient No. L | Lab. test | Cycle | Examination date | N | Std. value | Normal<br>range | NCI-<br>CTCAE<br>V4.03 grade |
|---|---|---|---|---|---|---|---|---|

Table 11.5.1. 4 Supportive listing: Patients with missing grade for hematological abnormalities

| Dose level | Patient No. Lab. test | Cycle | Examination date | N | Std. value | Normal<br>range | NCI-<br>CTCAE<br>V4.03 grade |
|---|---|---|---|---|---|---|---|

#### 11.5.2. Biochemical abnormalities

Table 11.5.2. 1 Biochemical abnormalities: Worst grade per patient DLn **Event** Grade 0 Grade 1 Grade 2 Grade 3 Grade 4 Grade 1-2 Grade 3-4 Grade 1-4 N AP increase ALT increase AST increase Amylase increase XXXXX Notes: Percentage is based on number of patients by dose level. Table 11.5.2. 2 Biochemical abnormalities: Worst grade per cycle **Event** DLnGrade 0 Grade 1 Grade 2 Grade 3 Grade 4 Grade 1-2 Grade 3-4 Grade 1-4 AP increase ALT increase AST increase Amylase increase XXXXX Notes: Percentage is based on number of patients by dose level. Supportive listing: Patients with grade ≥3 biochemical abnormalities NCI-Value **CTCAE** Dose level Patient No.Lab. test Cycle Examination date N Std. value (xULN) V4.03 grade Table 11.5.2. 4 Supportive listing: Patients with missing grade for biochemical abnormalities NCI-Value Dose level Patient No.Lab. test Cycle Examination date N Std. value CTCAE (xULN) V4.03 grade

# 11.5.3. Laboratory Values over Time

Table 11.5.3. 1 Shift of hematological abnormalities. Baseline grade vs worst grade on treatment

| Table 11.5.3. | 1 Shift of hematological abnormalities | | Wo | orst g | grade | ont | reatr | nent | | . 1 |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Baseline grade | Gr.<br>N | | Gr | | Gr. | | Gr | |
| DLI | Anemia | 0 | 11 | 70 | IN | 70 | IN | 70 | 11 | 70 |
| | | 4 | | | | | | | | |
| | Leukopenia | 0 | | | | | | | | |
| | | 4 | | | | | | | | |
| | _ | 0 | | | | | | | | |
| | | 4 | | | | | | | | |
| | Anemia | 0 | | | | | | | | |
| | | 4 | | | | | | | | |
| | Leukopenia | 0 | | | | | | | | |
| | _ | | | | | | | | | |
| | | 4 | | | | | | | | |
| | _ | 0 | | | | | | | | |
| | | 4 | | | | | | | | |
| DLn | Anemia | 0 | | | | | | | | |
| | Leukopenia | 4<br>0 | | | | | | | | |
| | Leukopenia | | | | | | | | | |
| | | 4 | | | | | | | | |
| | <del>_</del> | 0 | | | | | | | | |
| All treated | Anemia | 0 | | | | | | | | |
| population | Allema | | | | | | | | | |
| ророжион | | 4 | | | | | | | | |
| | Leukopenia | 0 | | | | | | | | |
| | _ | 4<br>0 | | | | | | | | |
| | | 4 | | | | | | | | |

Table 11.5.3. 2 Shift of biochemical abnormalities. Baseline grade vs worst grade on treatment

| Table 11.5.3. 2 Sh | int of biochemical | abnormalities. Basel | | | e on trea | | on u | caume | Ш | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Baseline grade | Gr.1 | | Gr. 2 | | Gr. 3 | 3 | Gr. 4 | Į. |
| | | Busemie grune | N | % | N | % | N | % | N | % |
| DLI | AP increase | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| | ALT increase | 0 | | | | | | | | |
| | | 4 | | | | | | | | |
| | ••• | 0 | | | | | | | | |
| | | ••• | | | | | | | | |
| | | 4 | | | | | | | | |
| ••• | AP increase | 0 | | | | | | | | |
| | | 4 | | | | | | | | |
| | ALT increase | 0 | | | | | | | | |
| | | 4 | | | | | | | | |
| | ••• | 0 | | | | | | | | |
| | | <br>4 | | | | | | | | |
| DLn | AP increase | 0 | | | | | | | | |
| DEII | 7 II IIRICIDO | | | | | | | | | |
| | | 4 | | | | | | | | |
| | ALT increase | 0 | | | | | | | | |
| | | 4<br>0 | | | | | | | | |
| | ••• | | | | | | | | | |
| | | 4 | | | | | | | | |
| All Treated Population | AP increase | 0 | | | | | | | | |
| | A.T. (T) . | 4 | | | | | | | | |
| | ALT increase | 0 | | | | | | | | |
| | | 4 | | | | | | | | |
| | ••• | 0 | | | | | | | | |
| | | 4 | | | | | | | | |

Table 11.5.3. 3 Worst severity of hematological abnormalities during the first and later cycles

| Overtime | Toxicity | DLI | DLII | DLIII | <br> | DL n |
|----------|-------------------|-----|------|-------|------|------|
| Cycle 1 | Anemia/ | | | | | |
| | Grade 1 - 4, n(%) | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Grade 4 | | | | | |
| Cycle>1 | Anemia/ | | | | | |
| - | Grade 1 - 4, n(%) | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Grade 4 | | | | | |

Notes: Percentage is based on number of patients by dose level.

Table 11.5.3. 4 Worst severity of biochemical abnormalities during the first and later cycles

| Overtime | Toxicity | DLI | DLII | DLIII | <br> | DL n |
|----------|-------------------|-----|------|-------|------|------|
| Cycle 1 | AP increase/ | | | | | |
| • | Grade 1 - 4, n(%) | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Grade 4 | | | | | |
| Cycle>1 | AP increase/ | | | | | |
| | Grade 1 - 4, n(%) | | | | | |
| | Grade 1 | | | | | |
| | Grade 2 | | | | | |
| | Grade 3 | | | | | |
| | Grade 4 | | | | | |

Notes: Percentage is based on number of patients by dose level.

Table 11.5.3. 5 Pattern of neutropenia/thrombocytopenia

| Dose level (X) | | | | | Day of | recover<br>x ULN | y to XX | Day | s to reco | overy |
|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory<br>abnomnalities<br>NEU (N=XX)<br>PLAT (N=XX) | Onset day grade 3/4 | Day of recovery<br>to grade 1 | Days<br>recovery | to | <=21 | 22-28 | >28 | <=15 | 16-24 | >=25 |

Table 11.5.3. 6 Pattern of hepatobiliary parameters

| - 110-10 - 1-10-10-1 | 1 44444111 01 114 | pure grand | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Dose level (X) | | | | Da | - | ecovery<br>ULN | to XX | Day | s to reco | overy |
| Laboratory<br>abnormalities<br>ALT (N=XX)<br>AST (N=XX) | Onset day grade 3/4 | Day of recovery to 3 x ULN | Days<br>recovery | to <=2 | 21 2 | 22-28 | >28 | <=15 | 16-24 | >=25 |

# 11.6. Other observation related to safety

# 11.6.1. Vital signs, physical findings and other observations related to safety

| | | Baseline | Cycle 1 | Cycle 2 | | Cycle N |
|---|---|---|---|---|---|---|
| ose level | Patient No. | PS | PS | PS | | PS |
| LI(N=XX | ) | | | | | |
| LII(N=XX | 7) | | | | | |
| | <b>L</b> ) | | | | | |
| DLN(N=XX | <u>()</u> | | | | | |
| L11(11 22 | 1) | | | | | |
| Table 11.6. | 1. 2 Physic | cal examination | n during the stud | y by cycle and d | ose level | |
| able 11.6. | 1.2 Physic | cal examination<br>Baseline | n during the stud<br>Cycle 1 | y by cycle and d<br>Cycle 2 | ose level | Cycle N |
| Dose level | Patient No. | | | | ose level<br><br>Physical exam | Cycle N Physical exam |
| Dose level | Patient No. | Baseline | Cycle 1 | Cycle 2 | | |
| Table 11.6. Dose level DLI(N=XX | Patient No. | Baseline | Cycle 1 | Cycle 2 | | |
| Oose level<br>DLI (N=XX | Patient No. | Baseline | Cycle 1 | Cycle 2 | | |
| Dose level | Patient No. | Baseline | Cycle 1 | Cycle 2 | | |
| Oose level<br>DLI (N=XX | Patient No. | Baseline | Cycle 1 | Cycle 2 | | |
| Oose level<br>DLI (N=XX | Patient No. | Baseline | Cycle 1 | Cycle 2 | | |
| Oose level DLI(N=XX DLII(N=XX | Patient No. | Baseline | Cycle 1 | Cycle 2 | | |
| Oose level DLI (N=XX DLII (N=XX | Patient No. | Baseline | Cycle 1 | Cycle 2 | | |

| Table 11.6 | .1.3 Weig | ght gain-loss during | the study by d | lose level | | |
|---|---|---|---|---|---|---|
| Dose level | Patient No. | Weight at baseline (kg) | Cycle 1 | Cycle 2 | | Cycle N |
| | | vveigna oasemie (ng) | % change | % change | % change | % change |
| DLI(N=X | X) | | | | | |
| DLII(N=X | X) | | | | | |
| DLII(IV-A | Λ) | | | | | |
| DL N (N | = | | | | | |
| XX) | | | | | | |
| | | | | • | • | |
| Гable 11.6 | .1.4 Vita | l sign (pulse) during | | | | |
| | | Baseline | Cycle 1 | Cycle 2 | | Cycle N |
| Dose level | Patient No | o. Pulse | Pulse | Pulse | Pulse | Pulse |
| DLI(N=X | X) | | | | | |
| DI HAL M | 30 | | | | | |
| DLII(N=X | X) | | | | | |
| DLN(N=X | (X) | | | | | _ |
| ` | , | | | | | |
| Γable 11.6 | 1.5 Vital | l sign (temperature) | during the stu | dy by cycle and | dose level | |
| 14010 11.0 | .1. 5 110 | | Cycle 1 | Cycle 2 | | Cycle N |
| Dose level | Patient No | | Temperature | Temperature | Temperature | Temperature |
| DLI(N=X | | 5. Temperature | Temperature | Terriperanie | Terriperature | Tomportunio |
| DE1(11 12 | ••) | | | | | |
| DLII(N=X | X) | | | | | , |
| * | * | | | | | |
| DLN(N=X | (X) | | | | | |

| | | Baseline | Cycle 1 | Cycle 2 | | Cycle N |
|---|---|---|---|---|---|---|
| Dose level | Patient No. | BPS | BPS | BPS | BPS | BPS |
| DLI(N=XX | () | | | | | |
| DLII(N=XX | X) | | | | | |
| DLN(N=X | X) | | | | | |
| | | | | • | | • |
| Гable 11.6. | 1. 7 Vital si | | | cycle and dose | | G 1 M |
| | | Baseline | Cycle 1 | Cycle 2 | | Cycle N |
| Dose level | Patient No. | BPD | BPD | BPD | BPD | BPD |
| DLI(N=XX | <b>(</b> ) | | | | | |
| DLII(N=XX | X) | | | | | |
| • • | | | | | | |
| DLN(N=X | X) | | | | | |
| Fabla 11 6 | 1 0 ECC 4 | uning the study | · h·· avala and d | laga laval | | |
| 1 4016 11.0. | 1. 0 ECU UL | Baseline | by cycle and d<br>Cycle 1 | Cycle 2 | | Cycle N |
| Dose level | Patient No. | ECG | ECG | ECG | ECG | ECG |
| DLI(N=XX | | | | | | |
| )LI(I\ 12) | <b>.</b> ) | | | | | |
| DLII(N=XX | <u> </u> | | | | | |
| | <del>*)</del> | | | | | |
| N NIAI-V | <b>V</b> ) | | | | | |
| DLN(N=X | X) | | | | | |

| | · | Baseline | Cycle 1 | e and dose level<br>Cycle2 | | Cycle N |
|---|---|---|---|---|---|---|
| Dose level | Patient No. | PRI | PRI | PRI | PRI | PRI |
| DLI(N=XX | <u>()</u> | | | | | |
| · | , | | | | | |
| DLII(N=X | X) | | | | | |
| DLN(N=X | X) | | | | | |
| P.1.1 11 C | 1 10 500 ( | ATIVA | | | | |
| abie 11.6. | 1. 10 ECG (C | Baseline | Cycle 1 | e and dose level<br>Cycle2 | | Cycle N |
| Dose level | Patient No. | QTI | QTI | QTI | QTI | QTI |
| DLI(N=XX | | <b>X</b> | <b>—</b> | <b>X</b> | <b>(</b> | <b>~</b> |
| )L1(1\ 7\) | <b>S</b> ) | | | | | |
| DLII(N=XX | X) | | | | | |
| 222(11) | -) | | | | | |
| DLN(N=X | X) | | | | | |
| · | | | | | | |
| | | | | • | | • |
| Table 11.6. | 1. 11 ECG (C | | | e and dose level | | ConlaN |
| . 1 1 | D.C. (M | Baseline | Cycle 1 | Cycle 2 | ОТ | Cycle N |
| Dose level | Patient No. | QTc | QTc | QTc | QTc | QTc |
| DLI(N=XX | 3) | | | | | |
| NI HAL M | | | | | | _ |
| DLII(N=X | X) | | | | | |
| N NIAI-N | <b>V</b> ) | | | | | |
| DLN(N=X | X) | | | | | |

Table 11.6.1. 12 ECG (VR) during the study by cycle and dose level Cycle N Baseline Cycle 1 Cycle 2 . . . Dose level VR Patient No. VR VR VR VR DLI(N=XX)  $\overline{DLII(N=XX)}$ ---DLN(N=XX)

## 11.7. Concomitant medication

## 11.7.1. Concomitant medication during study

Table 11.7.1. 1 Concomitant medication during study (ATC 1 and 4) by dose level

| | | <u> </u> | \ | | 2 | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Medication Term | Medication Term | Medication Term | DLI | | DLII | | DLIII | | | | | | DL n | | Total | |
| (ATC level 1) | (ATC level 2) | (ATC level 4) | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

Notes: Percentage is based on number of patients by dose level.

Table 11.7.1. 2 Transfusions / EPO (Patients with transfusions and/or EPO)

| Medication Term | Medication Term | Medication Term | DLI | | DLII | | DLIII | | | | | | DL n | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (ATC level 1) | (ATC level 2) | (ATC level 4) | N | % | N | % | N | % | N | % | N | % | N | % | N | % |

Platelet transfusion

RBC transfusion

EPO

. . .

## 12. APPENDIX III. EFFICACY EVALUATION

## 12.1. Efficacy analysis

All efficacy tables and graphs will be split by type of evaluation criteria, if appropriate, and any group of interest will be adequately represented as shown in Table 12.1.1.1. Otherwise, listings with individual patient responses will be produced and additional details for patients responding or showing stabilizations  $\geq 4$  months will be provided.

## **12.1.1.** Response

Table 12.1.1. 1 Overall response by dose level. Treated patients

| Or rowall mornousco | DL: | DLI | | DLII | | DLIII | | | | | DL n | | Tota | 1 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Overall response | N | % | N | % | N | % | N | % | N | % | N | % | N | % |
| CR | | | | | | | | | | | | | | |
| PR | | | | | | | | | | | | | | |
| SD<4 months | | | | | | | | | | | | | | |
| SD≥4 months | | | | | | | | | | | | | | |
| PD | | | | | | | | | | | | | | |
| NE | | | | | | | | | | | | | | |
| Total | | | | | | | | | | | | | | |

Notes: Percentage is based on number of patients by dose level.

Table 12.1.1. 2 Overall response by dose level. Evaluable patients

| DL1 | DLI | | DLII | | DLIII | | | | | | DL n | | 1 |
|-----|-----|---|------|---|-------|---|---|---|---|---|------|---|---|
| N | % | N | % | N | % | N | % | N | % | N | % | N | % |
| | | | | | | | | | | | - | | |

Table 12.1.1. 3 Tumor marker evolution during the study

| | | | Baseline | Cycle 1 | |
|---|---|---|---|---|---|
| Dose<br>level | Patient<br>No. | Tumor<br>type/Tumor<br>marker | Value | Value | Best change Time to best during change during treatment (%) treatment |
| I | | | | | |
| N | | | | | |

<sup>\*</sup> Patients not qualifying for response or progression disease.

#### Table 12.1.1. 4 Progression-free survival. Treated population

Summary

N=XX

Events X(XX.X%)

Censored X (XXXX%)

Median X.X 95% CI (X.X-X.X)

PFS at 3 months XX.X% 95% CI XX.XX%-XX.X%)

PFS at 6 months XX.X% 95% CI XX.XX%-XX.X%)

#### Table 12.1.1. 5 Progression-free survival. Evaluable population

Summary

N=XX

Events X(XXX%)

Censored X (XXXX%)

Median X.X 95% CI (X.X-X.X)

PFS at 3 months XX.X% 95% CI XX.XX%-XX.X%)

PFS at 6 months XXXX% 95% CIXXXXX%-XXXX%)

#### Table 12.1.1. 6 Duration of response

Summary

N=XX

Events X(XX.X%)

Censored X (XXXX%)

Median X.X 95% CI (X.X-X.X)

Duration of response at 3 months XX.X% 95% CI XX.XX%-XX.X%)

Duration of response at 6 months XX.X% 95% CI XX.XX%-XX.X%)

| Table 12.1.1. 7 | Characteristics of | natients with | evidence of | clinical benefit* |
|---|---|---|---|---|

| Dose level | Patient No. Gender Age I | PS | No. of Tumor typelines of previous (previous CT) | Best response previous CT | toTTP previous received CT (months) PM060184 | Overall response | PFS<br>(months) | Reason for treatment Cause of death discontinuation |
|---|---|---|---|---|---|---|---|---|
| | | | CI | _ | PIVIU0U184 | _ | | |

(\*) "Evidence of clinical benefit" is defined as response (CR, PR) or SD>4 months and/or no evidence of PD with decreasing tumor markers, if not evaluable per RECIST.

Table 12.1.1. 8 Supportive listing: efficacy dataset analyzed

| Dose level | Patient No. | Tumortype | Evaluable | Evaluation criteria | Best response | Progression | Progression date | Death | Death date |
|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|

# 13. FIGURES

# 13.1. Hematological profile

Figure 13.1. 1 Pattern of hematological/non-hematological DLTs in individual patients



### 13.2. Transaminase Profile

Figure 13.2. 1 Transaminase series. Patient XX



Figure 13.2. 2 Bar charts of hematological/biochemical laboratory abnormalities by dose level



Figure 13.2. 3 Hematology / Transaminase. Worst severity by cycle



# 13.3. Time to event graphs

Figure 13.3. 1 Progression-free survival (PFS)

Progression Free Survival (PFS)



Median 1.6 95% CI (1.0-2.7)
PFS at 3 months 21.2% 95% CI (3.9%-38.4%)
PFS at 6 months 5.3% 95% CI (0%-15.3%)
PFS at 12 months 5.3% 95% CI (0%-15.3%)

### 14. DATABASE LISTINGS

- Listing 14.1 Patient registration
- Listing 14.2 Demography
- Listing 14.3 Birth control and pregnancy test
- Listing 14.4 Relevant prior history
- Listing 14.5 Cancer history
- Listing 14.6 Prior surgery
- Listing 14.7 Prior radiotherapy
- Listing 14.8 Prior anticancer therapy
- Listing 14.9 Drug administration
- Listing 14.10 End of treatment
- Listing 14.11 Adverse events
- Listing 14.12.1 Hematology
- Listing 14.12.2 Serum biochemistry
- Listing 14.12.3 Coagulogram
- Listing 14.12.4 Other tests
- Listing 14.13 Physical examination
- Listing 14.14 Performance status (PS)
- Listing 14.15 Vital signs
- Listing 14.16 Electrocardiogram
- Listing 14.17 Left ventricular ejection fraction (LVEF) results
- Listing 14.18 Concomitant therapy
- Listing 14.19 Tumor assessment
- Listing 14.20 Tumor response cycles
- Listing 14.21 Clinical response cycles
- Listing 14.22 Best response
- Listing 14.23 Summary efficacy
- Listing 14.24 Follow-up status
- Listing 14.25 Follow-up: Antitumor therapy
- Listing 14.26 Death report
- Listing 14.27 Off study
- Listing 14.28 Signature report